### Statistical Analysis Plan

Protocol Number: MT-7117-G01

A Phase 3, Multicenter, Randomized, Double-Blind,
Placebo-Controlled Study to Evaluate Efficacy, Safety,
and Tolerability of MT-7117 in Adults and Adolescents
With Erythropoietic Protoporphyria or X-Linked
Protoporphyria

Version Number: 3.0 Date: 16 Sep 2022

NCT number: NCT04402489

## Statistical Analysis Plan

#### Protocol No. MT-7117-G01

A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Efficacy, Safety, and Tolerability of MT-7117 in Adults and Adolescents with Erythropoietic Protoporphyria or X-Linked Protoporphyria

| Prepared By: | Mitsubishi Tanabe Pharma Development America |
|--------------|----------------------------------------------|
| Version: | V3.0 |
| Date: | 16SEP2022 |

### APPROVAL FORM

### Statistical Analysis Plan

| Protocol No. | MT-7117-G01 |
|---|---|
| Protocol Title | A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-<br>Controlled Study to Evaluate Efficacy, Safety, and Tolerability of |
| | MT-7117 in Adults and Adolescents with Erythropoietic |
| | Protoporphyria or X-Linked Protoporphyria |
| Version / Date | v3.0/ 16SEP2022 |

#### Authors:

| Statistics Author | |
|----------------------|---------------|
| Print Name: | |
| Position: | |
| Print Name: | |
| Position: | |
| Clinical Pharmacokir | netics Author |
| Print Name: | |
| Position: | |

Approved by:

| Statistic Approver | |
|--------------------|------------------|
| Print Name: | |
| Position: | Responsible STAT |
| Signature: | |
| Approval date: | |
| Clinical Pharmaco | kinetic Approver |
| Print Name: | |
| Position: | Responsible CP |
| Signature: | |
| Approval date: | |

### TABLE OF CONTENTS

| STA | TIST | TCAL ANALYSIS PLAN | . 1 |
|---|---|---|---|
| APP | ROV | AL FORM | . 2 |
| TAB | LE ( | OF CONTENTS | . 4 |
| ABE | BREV | /IATIONS | . 7 |
| 1 | INT | RODUCTION | . 8 |
| 2 | STU | DY OBJECTIVE AND ENDPOINTS | . 8 |
| | <ul><li>2.1</li><li>2.2</li><li>2.3</li></ul> | Study Objectives Estimand 2.2.1 Primary estimand 2.2.2 Secondary Estimand Study Endpoints 2.3.1 Primary Efficacy Endpoint for Primary Week26 (DBT) data analysis 2.3.2 Secondary Efficacy Endpoints for Primary Week26 (DBT) Data Analysis | .9<br>.9<br>10<br>10<br>11<br>12<br>13 |
| | C.T. | 2.3.7 Pharmacogenetics Assessments | |
| 3 | STU | DY DESIGN | Į <b>4</b> |
| | <ul><li>3.1</li><li>3.2</li><li>3.3</li></ul> | Study Design | 16<br>20<br>20 |
| 4 | PLA | NNED ANALYSIS2 | 21 |
| | 4.1<br>4.2 | Primary Week 26 Analysis | |
| 5 | ANA | ALYSIS POPULATIONS2 | 22 |
| | 5.1<br>5.2<br>5.3<br>5.4 | Randomized (RAND) Population | 22<br>22 |
| 6 | STA | TISTICAL CONSIDERATIONS | 23 |
| | 6.1 | Descriptive Statistics | 23 |

| | 6.2 | Statistica | l Tests | . 23 |
|---|---|---|---|---|
| | 6.3 | Stratifica | tion registration errors | . 23 |
| | 6.4 | Dosing st | uspension | . 24 |
| 7 | DA | A CONVI | ENTIONS | . 24 |
| | 7.1 | Treatmen | nt Group Definitions and The Corresponding Analyzed Period Data | . 24 |
| | 7.2 | Analysis | Variable Definitions | . 25 |
| | | 7.2.1 St | udy Subjects | . 25 |
| | | 7.2.1 | .1 Protocol Deviation | . 25 |
| | | 7.2.1 | .2 Demographic and Other Baseline Characteristics | . 25 |
| | | | 1.3 Medical Ĥistory | |
| | | | .4 Prior or Concomitant Medication | |
| | | | .5 Treatment Duration and Compliance | |
| | | | fficacy assessments | |
| | | 7.2.2 | 2.1 The Sunrise and Sunset Time to Use | .27 |
| | | | 2.2 Data Handling of eDiary records | |
| | | | 2.3 Derivation Rule for Efficacy Endpoints from eDiary records | |
| | | | 2.4 PGIC 31 | |
| | | | 2.5 PGIS 32 | |
| | | | 2.6 PROMIS-5732 | |
| | | | afety Assessments | 33 |
| | | 7.2.3 | 3.1 Adverse Events | 33 |
| | | | 3.2 Physical examiniation | |
| | | | 3.3 Laboratory Tests | |
| | | | 3.4 12-Lead ECG | |
| | | | ata Handling of PK data and melanin density data | |
| | 7.3 | | Visit Definitions | |
| | 7.3<br>7.4 | • | Idling Convention for Missing Data | |
| | 7.4 | <b>Да</b> іа Пап | diling Convention for Missing Data | , 37 |
| 8 | STA | TISTICAL | METHODOLOGY | . 39 |
| | 8.1 | Study Sul | bjects | . 39 |
| | | | ubject Disposition | |
| | | 8.1.2 Aı | nalysis Populations | . 39 |
| | | 8.1.3 Pr | otocol Deviations | . 39 |
| | | 8.1.4 St | ratification Registration Errors | . 39 |
| | | | emographic and Other Baseline Characteristics | |
| | | | edical History | |
| | | | ior or Concomitant Medications | |
| | | | ohibited medication | |
| | | | reatment Duration and Compliance | |
| | | | tzpatrick skin scale test | |
| | | | ubject Questionnaire for Study Medication | |
| | 8.2 | | Assessments | |
| | 0.2 | • | imary Efficacy Endpoint | |
| | | | econdary Efficacy Endpoints | |
| | | | sploratory Efficacy Endpoints | |
| | 0 2 | | | |
| | 8.3 | Salety As | ssessments | . J4 |

| Stat<br>Prot | istical .<br>ocol N | Analysis<br>o. MT-7 | Plan<br>117-G01 | Mitsubishi Tanabe Pharma Development America |
|---|---|---|---|---|
| | 8.4<br>8.5 | 8.3.1<br>8.3.2<br>8.3.3<br>8.3.4<br>8.3.5<br>8.3.6<br>Pharm | Adverse Events Laboratory Tests Vital Signs | |
| 9 | 8.6<br>DAT | _ | | |
| | 9.1<br>9.2<br>9.3 | Numb<br>Treatr | per of Digits to Report<br>nent Groups to Report | |
| 10 | CH | ANGE | FROM THE PROTOCOL | 63 |
| 11 | SOF | TWAR | E | 64 |
| 12 | REF | EREN | CES | 64 |
| 13 | | | | 64 |
| 14 | APF | ENDE | ζ | 67 |
| | 14.2 | S | MQ List of Hepatic TEAE in Med | DRA version 23.173 |
| | | | LIST OF TA | BLES |
| | | | • | 16 |
| | | | | 17 |
| TAI | BLE 2 | ANAI | LYSIS VISIT WINDOW FOR DIA | RY DATA35 |
| TAI | BLE 3 | ANAI | YSIS VISIT WINDOW FOR NO | N-DIARY DATA36 |

### **ABBREVIATIONS**

| Abbreviations | Definitions |
|---------------|-------------------------------------------------|
| AE | adverse event |
| ALT | alanine transaminase |
| ALP | alkaline phosphatase |
| ANCOVA | analysis of covariance |
| AST | aspartate transaminase |
| ATC | anatomical therapeutic chemical |
| BDR | blinded data review |
| BMI | body mass index |
| CI | confidence interval |
| DBE | double-blind extension |
| DBT | double-blind treatment |
| DP | decimal places |
| ECG | electrocardiogram |
| EPP | Erythropoietic protoporphyria |
| FAS | full analysis set |
| ITT | intent-to-treat |
| MedDRA | medical dictionary for regulatory activities |
| MMRM | mixed model repeated measures |
| PD | pharmacodynamics |
| PK | pharmacokinetics |
| PT | preferred term |
| QTcB | Corrected QT interval using Bazett's formula |
| QTcF | Corrected QT interval using Fredrecia's formula |
| SAP | statistical analysis plan |
| SAE | serious adverse event |
| SAF | safety population |
| SD | standard deviation |
| SOC | system organ class |
| TEAE | treatment emergent adverse event |
| TESAE | treatment emergent serious adverse events |
| ULN | upper limit of normal range |
| WHO | World Health Organization |
| XLP | X linked porphyria |

#### 1 INTRODUCTION

This statistical analysis plan (SAP) is based on the final global master protocol version 4.1 dated 9AUG2021, the final Japan specific protocol (v4.2) dated 24 August 2021, and the final Norway specific protocol (v4.3) dated 24 August 2021, and the final Germany specific protocol (v4.4) dated 24 August 2021 and , and the final Canada specific protocol (v4.5) dated 24 August 2021. The plan covers statistical analysis, tabulations, and listings of the study data to assess the efficacy, safety, and PK of and doses of MT-7117 compared to placebo. Any statistical analysis details described in this document supersede any description of statistical analysis in the protocol.

The SAP is prepared by MTDA and MTPC data science and reviewed by MTDA clinical study team and MTPC data science following GLB-BST-SOP002 ver.7. The statistical analyses and production of the outputs described in the SAP will be conducted and QCed by using SAS version 9.4 or higher. The final analyses and outputs will be approved by MTPC/MTDA Data Science.

This SAP has been approved and signed as Version 1.0 and Version 1.1 for FDA SAP communication. Version 2.0 will be finalized for the Primary Week 26 analysis prior to Week 26 database lock, and Version 3.0 will be finalized for the final analysis prior to the final database lock.

The analysis plan for the PPKPD will be described in a separate document and the results will be separately reported.

For the qualitative exit interview questionnaire, the analysis plan, the dataset and the results will be separately created and reported.

#### 2 STUDY OBJECTIVE AND ENDPOINTS

#### 2.1 Study Objectives

#### **Primary:**

- To investigate the efficacy of MT-7117 on time to onset and severity of first prodromal symptoms (burning, tingling, itching, or stinging) associated with sunlight exposure in adults and adolescents with EPP or XLP.

#### Secondary:

- To investigate the effect on patient-reported quality of life in adults and adolescents with EPP or XLP.
- To investigate the effect on the percentage of responders based on the within-subject meaningful threshold for time to first prodromal symptom in adults and adolescents with EPP or XLP.

- To investigate the effect on number and severity of sunlight-induced pain events (prodrome and phototoxic reactions) in adults and adolescents with EPP or XLP.

#### **Exploratory:**

- To investigate the effect on sunlight exposure duration in adults and adolescents with EPP or XLP.
- To investigate the effect on melanin density in adults and adolescents with EPP or XLP.
- To investigate the PK/pharmacodynamic (PD) relationship in adults and adolescents with EPP or XLP.

#### Safety:

- To assess the long-term safety and tolerability of MT-7117.

#### 2.2 Estimand

#### 2.2.1 Primary estimand

The primary estimand construction elements for this study are:

- Population: All randomized subjects who received at least 1 dose of study medication with baseline and post-randomization sunlight exposure diary assessment.
- Variable: Change from baseline in average daily sunlight exposure time (minutes) to first prodromal symptom associated with sunlight exposure between 1 hour post sunrise and 1 hour pre-sunset at Week 26 (Visit 7).
- Inter-current event of treatment discontinuation using treatment policy: Regardless of early discontinuation of study drug due to any reason until the end of the double-blind treatment period.
- Population-level summary: Absolute mean difference in change from baseline in average daily sunlight exposure time (minutes) to first prodromal symptom between MT-7117 and placebo groups.

The primary estimand will be based on effectiveness assumption (de-facto) using treatment policy: The treatment effect will be attributable to the subject's initially randomized treatment regardless of treatment discontinuation.

#### 2.2.2 Secondary Estimand

The secondary estimand construction elements to be tested as supportive analysis for this study are:

- Population: All randomized subjects who received at least 1 dose of study medication with baseline and post-randomization sunlight exposure diary assessment.
- Variable: Change from baseline in average daily sunlight exposure time (minutes) to first prodromal symptom associated with sunlight exposure between 1 hour post sunrise and

- 1 hour pre-sunset at Week 26 (Visit 7).
- Inter-current event of treatment discontinuation using hypothetical strategy: If subjects could have treatment completion until the end of the double-blind treatment period.
- Population-level summary: Absolute mean difference in change from baseline in average daily sunlight exposure time (minutes) to first prodromal symptom between MT-7117 and placebo groups.

The secondary estimand will be based on efficacy assumption (de-jure) using a hypothetical strategy: The treatment effect will be attributable to the subject's initially randomized treatment if subjects could have stayed on study until the end of the double-blind treatment period.

#### 2.3 Study Endpoints

#### 2.3.1 Primary Efficacy Endpoint for Primary Week26 (DBT) data analysis

• Change from baseline in average daily sunlight exposure time (minutes) to first prodromal symptom (burning, tingling, itching, or stinging) associated with sunlight exposure between 1 hour post sunrise and 1 hour pre-sunset at Week 26 (Visit 7).

To calculate the average daily sunlight exposure time to first prodromal symptom, a 14 day window on or before a timepoint (Week 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, and 26) will be used. For baseline, a 14 day window before Day 1 will be used. A 14 day window will be applied to similar situations for other efficacy endpoints related to sunlight exposure diary.

#### 2.3.2 Secondary Efficacy Endpoints for Primary Week26 (DBT) Data Analysis

- Patient Global Impression of Change (PGIC) at Week 26.
- Total number of sunlight-induced pain events defined as prodromal symptoms (burning, tingling, itching, or stinging) with pain rating of 1-10 on the Likert scale during the 26-week double-blind treatment period.
- Change from baseline for total score in the domain of pain intensity in the PROMIS-57 at Week 26.
- The percentage of subjects who are responders based on average daily sunlight exposure time to first prodromal symptom associated with sunlight exposure between 1 hour post sunrise and 1 hour pre-sunset defined by within-subject meaningful change of 66 minutes increase from baseline to Week 26.
- Change from baseline for total score in the domain of physical function in the PROMIS-57 at Week 26.

#### 2.3.3 Exploratory Efficacy Endpoints for Primary Week26 (DBT) Data Analysis

- Change from baseline for in-clinic sunlight exposure time (minutes) to the first prodromal symptoms or end of test, whichever comes first.
- Total time (hours) during the 26-week double-blind treatment period in duration of sunlight exposure between 1 hour post sunrise and 1 hour pre-sunset without prodromal symptoms.
- Total time (hours) during the 26-week double-blind treatment period in duration of sunlight exposure between 1 hour post sunrise and 1 hour pre-sunset without prodromal symptom with the severity of greater than 0 on 11-point Likert scale and without phototoxic reactions (pain-free time hours).
- Change from baseline in the average daily mean intensity on an 11-point Likert scale of the subject's prodromal symptoms over time during the 26-week double-blind treatment period.
- Change from baseline in average daily duration (minutes) of prodromal symptoms during the 26-week double-blind treatment period.
- Total number of sunlight-induced pain events defined as phototoxic events during the 26-week double-blind treatment period.
- Total number of sunlight-induced non-prodrome, phototoxic reactions during the 26-week double-blind treatment period.
- Change from baseline in the average daily mean intensity of the subject's phototoxic reactions (associated with sun exposure) during the 26-week double-blind treatment period on an 11-point Likert scale.
- Change from baseline in average daily duration (minutes) of phototoxic reactions (associated with sun exposure) during the 26-week double-blind treatment period.
- Change from baseline and % change from baseline in melanin density at each visit by skin segments. Average of 6 skin segments for the change from baseline and % change from baseline in melanin density at each visit.
- Total number of days subject is exposed to sunlight for any duration without prodromal symptoms during the 26-week double-blind treatment period.
- Total number of days subject is exposed to sunlight for any duration without prodromal symptom with the severity of greater than 0 on 11-point Likert scale and without phototoxic reactions (pain-free days) during the 26-week double-blind treatment period.
- Change from baseline in average daily duration of sunlight exposure regardless of time of day without prodromal symptoms assessed at Week 26.
- Change from baseline for all total score and total score in each domain of, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, and pain interference in the PROMIS-57

- Change from baseline in Patient Global Impression of Severity (PGIS) at each visit.
- The percentage of subjects who are responders at Week 26 based on PGIC (Very Much Improved or Much Improved).
- Qualitative exit interview questionnaire about QoL at Week 26.
- Total number of days subjects went outdoors during the 26-week double-blind treatment period.
- Maximum and total severity of phototoxic reaction on an 11-point Likert scale.

#### 2.3.4 Exploratory Efficacy Endpoint for Double Blind Extention (DBE) Data Analysis

- Change from baseline in average daily sunlight exposure time (minutes) to first prodromal symptom (burning, tingling, itching, or stinging) associated with sunlight exposure between 1 hour post sunrise and 1 hour pre-sunset at each timepoint.
- Patient Global Impression of Change (PGIC) at each visit.
- Total number of sunlight-induced pain events defined as prodromal symptoms (burning, tingling, itching, or stinging) with pain rating of 1-10 on the Likert scale during each 26-week double-blind extention treatment.
- Change from baseline for all total score and total score in each domain the PROMIS-57 at each visit.
- The percentage of subjects who are responders based on average daily sunlight exposure time to first prodromal symptom associated with sunlight exposure between 1 hour post sunrise and 1 hour pre-sunset defined by within-subject meaningful change of 66 minutes increase from baseline at each time point.
- Change from baseline for in-clinic sunlight exposure time (minutes) to the first prodromal symptoms or end of test, whichever comes first.
- Total time (hours) during the 26-week double-blind extention period in duration of sunlight exposure between 1 hour post sunrise and 1 hour pre-sunset without prodromal symptoms.
- Total time (hours) during the 26-week double-blind extention period in duration of sunlight exposure between 1 hour post sunrise and 1 hour pre-sunset without prodromal symptom with the severity of greater than 0 on an 11-point Likert scale and without phototoxic reactions (pain-free time hours).
- Change from baseline in the average daily mean intensity on an 11-point Likert scale of the subject's prodromal symptoms over time during the 26-week double-blind extention period.

- Change from baseline in average daily duration (minutes) of prodromal symptoms during the 26-week double-blind extention period
- Total number of sunlight-induced pain events defined as phototoxic events during the 26week double-blind extention period
- Total number of sunlight-induced non-prodrome, phototoxic reactions during the 26-week double-blind extention period.
- Change from baseline in the average daily mean intensity of the subject's phototoxic reactions (associated with sun exposure) during the 26-week double-blind extention period on an 11-point Likert scale.
- Change from baseline in average daily duration (minutes) of phototoxic reactions (associated with sun exposure) during the 26-week double-blind extention period.
- Change from baseline and % change from baseline in melanin density at each visit by skin segments. Average of 6 skin segments for the change from baseline and % change from baseline in melanin density at each visit.
- Total number of days subject is exposed to sunlight for any duration between 1 hour post sunrise and 1 hour pre-sunset without prodromal symptoms during the 26-week double-blind extention period
- Total number of days subject is exposed to sunlight for any duration between 1 hour post sunrise and 1 hour pre-sunset without prodromal symptom with the severity of greater than 0 on an 11-point Likert scale and without phototoxic reactions (pain-free days) during the 26-week double-blind extention period
- Change from baseline in average daily duration of sunlight exposure regardless of time of day without prodromal symptoms assessed at each timepoint.
- Total number of days subjects went outdoors during the 26-week double-blind extention period
- Change from baseline in Patient Global Impression of Severity (PGIS) at each visit.
- The percentage of subjects who are responders at Week 52 based on PGIC (Very Much Improved or Much Improved).
- Maximum and total severity of phototoxic reaction on an 11-point Likert scale.

#### 2.3.5 Safety Endpoints

- Treatment-emergent adverse events (AEs) (including serious adverse events [SAEs] and adverse events of special interest [AESIs]).
- Physical examination.

- Vital signs (blood pressure, respiratory rate, pulse rate, body temperature and body weight).
- Clinical laboratory examinations (hematology, coagulation, biochemistry, and urinalysis), including liver function markers (ALT, AST, GGT, ALP, direct and total bilirubin).
- 12-lead ECG at Baseline and EOT.
- Nevi appearance (assessed by a dermatologist or other qualified site staff). Any nevi undergoing change of clinical concern during active treatment will be biopsied for follow up and evaluated by the central pathology lab.

#### 2.3.6 Pharmacokinetics Assessment(s)

 Assessment of plasma PK: Plasma concentrations of MT-7117 will be measured at protocol scheduled visits.

#### 2.3.7 Pharmacogenetics Assessments

#### 3 STUDY DESIGN

#### 3.1 Study Design

This is a Phase 3, randomized, double-blind, placebo-controlled study to assess the efficacy, tolerability, and safety of MT-7117 in adults and adolescents with EPP or XLP. The study consists of a 6-week screening period, a 26-week double-blind treatment period, an optional 26-week double-blinded extension (DBE) period, and a 6-week follow-up period at Week 58 (or Week 32 if DBE is not elected). The total participation period is approximately 64 weeks.

The study design is illustrated in Figure 1.

Subjects will attend the screening visit (Visit 1) up to 6 weeks before Randomization (Visit 2), in order to confirm eligibility and obtain pre-study safety assessments including nevi evaluation. Subjects will also be instructed how to use an electronic sunlight exposure diary (SED).

| At Visit 2, | |
|-------------|----------------------------------------|
| | , or placebo in a double-blind manner. |

The first dose will be administered at Visit 2 following baseline assessments including an inclinic sunlight exposure test at any time before randomization (Visit 1 or 2), and melanin density determination before randomization (Visit 2). Active or placebo will be administered once daily in the morning with or without food.

Subjects will subsequently attend in-clinic visits at Weeks 4 and 12 (Visits 4 and 6, respectively) during which assessments will be performed. In addition, subjects may undergo mobile laboratory or in-clinic visits for sample collection at Weeks 2 and 8 (Visits 3 and 5, respectively) to measure liver function markers (AST, ALT, GGT, ALP, direct and total bilirubin).

Subjects will attend the end of treatment visit at Week 26 or early termination visit (Visit 7 or Visit 11).

PK will be collected at scheduled visits for  $\ge 18$  to  $\le 75$ -year-olds. For  $\ge 12$  to  $\le 17$ -year-old subjects, a total of 9 PK samples at 3 time points will be collected: Day 1 (Visit 2) at 2, 4, 6, and 8 hours post-dose, Week 12 (Visit 6) at pre-dose and 3 hours post-dose, and Week 26 (Visit 7) at pre-dose and 2, and 4 hours post-dose.

Subjects will be offered participation in a 6-month extension where all participants are on active drug but are double-blinded to dose starting immediately after the end of the 26-week doubleblind treatment period. If study subjects elect to participate in the 26-week DBE after end of Visit 7 (EOT/Rand), subjects will remain blinded and subjects will be re-randomized. Subjects that received MT-7117 during the blinded period will continue the DBE in the same treatment arm and remain blinded. Subjects that received placebo will be randomized to receive

MT-7117 or in 1:1 ratio for the 26 weeks DBE period. the dose will be administered without re-randomization.

During the DBE, subjects will attend an in-clinic visit at Week 39 (Visit 10) where measurements will be performed. In addition, subjects may undergo mobile laboratory or inclinic visits for sample collection at Weeks 28 and 32 (Visits 8 and 9, respectively) to measure liver function markers (AST, ALT, GGT, ALP, direct and total bilirubin).

Subjects will attend the end of treatment visit at Week 52 or early termination visit (Visit 11). Following the last treatment visit, subjects will attend a follow-up visit at Week 58 (Week 32 if DBE is not elected) or 6 weeks after early termination visit.

Subjects who are permanently withdrawn from study drug early should be encouraged to continue in the study and complete all other study assessments without receiving study drug. If a patient decides to completely withdraw consent/assent from the study, every attempt should be made to have the patient complete an early termination visit (Visit 7 or Visit 11).



Figure 1 Study Design Schematic

#### 3.2 Schedule of Study Procedures

Study assessments and corresponding event schedules are summarized in the time and events schedule. The schedule of assessment in the global master protocol is shown in Table 1. The schedules of assessment for each country specific (Japan, Norway, Germany and Canada) are referred to each country specific protocol.

Mitsubishi Tanabe Pharma Development America

Table 1 Schedule of Assessments

Statistical Analysis Plan Protocol No. MT-7117-G01

| Study Period | Screenin | | Dou | Double-blind Treatment | Treatm | ent | | | Double-blind Extension | nd Extensio | | Follow-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Number | Visit 1 | Visit 2<br>(Random<br>ization) | Visit<br>3£ | Visit 4 | Visit | Visit 6 | Visit 7E (EOT/ Rand) | Visit 88 | Visit 95 | Visit 10 | Visit 11 <sup>a</sup><br>(EOT/<br>DBE) | Visit 12 <sup>£</sup> (EOS) |
| Study Week | Week -6 to<br>Week 0 | | Week<br>2 | Week<br>4 | Week<br>8 | Week<br>12 | Week<br>26 | Week<br>28 | Week<br>32 | Week<br>39 | Week<br>52 | Week<br>32 or 58 |
| Study Day ±<br>Window | Day -42 to<br>Study Day <sup>a</sup> | Day<br>1 | Day<br>14±5 | Day<br>29±7 | Day<br>57±7 | Day<br>85±7 | Day<br>183±7 | <b>Day</b><br>197±7 | <b>Day</b><br>225±7 | Day<br>274±7 | Day<br>365±7 | Day<br>407±7 |
| Informed<br>consent/assent <sup>b</sup> | × | | | | | | | | | | | |
| Inclusion/exclusion | × | × | | | | | | | | | | |
| Demographics | × | | | | | | | | | | | |
| Medical history | × | × | | | | | | | | | | |
| Randomization | | × | | | | | Xį | | | | | |
| Body weight | X | X | | X | | X | X | | | X | X | X |
| Height | X | | | | | | | | | | | |
| Physical examination <sup>c</sup> | × | X | * · | × | | X | X | | | X | X | × |
| Vital signs <sup>d</sup> | × | X | | X | | X | X | | | X | X | × |
| 12-lead ECG | X | | | | | | X | | | | X | |
| Hematology/coagul ation, biochemistry & urinalysis <sup>g</sup> | × | X | яX | X | 9X | X | X | <b>)X</b> | sX. | X | X | × |
| Blood collection for porphyrin and protoporphyrin levelsh | × | | | × | | X | X | | | × | × | |
| Fitzpatrick skin type | X | | | × | | × | × | | | X | X | |


Confidential

| Jan | 17-G01 |
|----------|--------------|
| lysis F | <b>AT-71</b> |
| al Ana | No. N |
| atistica | otocol |
| ឆ | 죠 |

| Protocol No. MT-7117-G01 | 11 | | | | | | 300 800 117 | Mitsubishi | Tanabe Pharr | Mitsubishi Tanabe Pharma Development America | ent America |
|---|---|---|---|---|---|---|---|---|---|---|---|
| assessment <sup>s</sup> | | | | | | | | | | | |
| Pregnancy test <sup>i</sup> | X | X | × | | × | × | | | × | × | × |
| PK sampling (blood) | | X | X | | × | × | | | X | X | |
| Blood sampling for PGx <sup>b</sup> | | X | | | | | | | | | |
| Dispensing of study medication | | X | X | | × | X | | | X | | |
| Medication<br>accountability | | | × | | X | X | | | X | X | |
| Subject Question<br>for study<br>medication <sup>k</sup> | | | , | | | X | | | | | |
| PROMIS-57 | | × | | | X | Х | | | X | × | X |
| PGIC | | | X | | | X | | | | X | |
| PGIS | | X | X | | X | X | Same and the second | | X | X | X |
| EOT/Exit interview questionnaire! | | | | | | X | | | | | |
| Sunlight exposure diaries <sup>m</sup> | | | | | | | | | | | $\uparrow$ |
| In-clinic sunlight exposure test <sup>a</sup> | | × | | | | × | | | | X | |
| Melanin density evaluation | | X | X | | × | X | | | | X | X |
| Nevi evaluation <sup>2</sup> | X | | X | 1987 · | X | X | | | X | X | X |
| Concomitant<br>medication | <b>\</b> | | | | | | | | | | <b>^</b> |
| Adverse events | <b> </b> | | | | | | | | | | 1 |

Abbreviations: DBE= double-blinded extension; ECG = electrocardiogram; EOS = end of study; EOT = end of treatment; PGIC = Patient Global Impression of Change; PGIS = Patient Global Impression of Severity; PGx = pharmacogenetics(s); PK = pharmacokinetic; PROMIS = Patient-Reported Outcomes Measurement Information System.

<sup>a</sup> A minimum of 7 days of outside exposure data is required prior to randomization.

b Blood samples will be collected for PGx analysis for those subjects who have specifically given informed consent/assent for optional PGx analysis at Visit 2.


Confidential

# Protocol No. MT-7117-G01 Statistical Analysis Plan

Mitsubishi Tanabe Pharma Development America

- c Complete physical examination will be performed at Visit 1 and an abbreviated physical examination will be performed at all other specified time points.
- <sup>1</sup> Vital signs include measurement of sitting blood pressure, respiratory rate, pulse rate, and body temperature.
- ECG will be assessed at Visit 7 for subjects who do not elect DBE. For subjects who elect DBE, ECG will be assessed at Visit 11.
- All study subjects who elect to participate in the 26-weeks DBE will be re-randomized. Subjects that received MT-7117 during the blinded period will continue the DBE in the same in 1:1 ratio for the 26 weeks DBE period. For subjects with or treatment arm and remain blinded. Subjects that received placebo will be randomized to receive MT-7117 dose will be administered without re-randomization. , the
- E At Visits 3, 5, 8, and 9, subjects may have mobile units or in-clinic visits to measure liver function markers (ALT, AST, GGT, ALP, direct and total bilirubin). Blood samples for liver function markers will be shipped to the central laboratory.
- Plasma total porphyrins and erythrocyte protoporphyrin will be assessed at Visits 1, 4, 6, 7, 10, and 11.
- For female subjects of child-bearing potential, a serum pregnancy test will be performed at Visit 1 and a urine pregnancy test will be performed at Visits 2, 4, 6, 7, 10, 11, and 12.
- For subjects who are  $\geq$ 18 to  $\leq$ 75: PK blood samples for MT-7117 will be collected and processed at Visit 2 (pre-dose), Visits 4, 6, 10, and 11 (any time), and Visit 7 (at the visit and 3 to 4 hours after the first PK sample collection [both post-dose]). Date and time of most recent dose, and date and time of PK sample collection will be recorded. Subjects who are >12 to <17 years old will have 9 PK samples at 3 time points collected. Visit 2 at 2, 4, 6, and 8 hours post-dose, Visit 6 at pre-dose and 3 hours post-dose, and Visit 7 at pre-dose and 2, and
- k Subjects will be asked whether they believe they received active or placebo treatment.
- <sup>1</sup> EOT/Exit interview will only be performed in selected countries.
- m Sunlight exposure data, presence of prodromal symptoms and sunlight-induced phototoxic reactions, their severity, and their onset/duration will be collected from Visits 1 through 12. Diary training will be performed at the first in-clinic visit during the screening period.
  - <sup>n</sup> In-clinic sunlight exposure test should be done once before randomization and once at Visit 7. For subjects who elect DBE, the test is also performed at Visit 11.
- o Nevi evaluation will be performed locally by a dermatologist or qualified site staff. Baseline nevi evaluation will be performed at any time during the Screening period before Randomization (Visit 1 or 2). The Nevi evaluation at Visit 12 is to assess for the reversibility if any suspicious nevi changes were observed during treatment as per the Investigator's (and/or dermatologist's or other qualified site staff) judgment. Any follow-up will be recorded in the eCRF. Nevi assessment will be described in a separate document.
- These assessments will be performed at Week 26 or early termination from the double-blind treatment period. If the visit is due to early termination, no double-blinded extension study medication is to be dispensed.
- <sup>q</sup> These assessments will be performed at Week 52 or early termination from the double-blinded extension period.
- All subjects will return to the study site for a 6-week follow-up visit at Week 58 (Week 32 if DBE is not elected) or 6 weeks after early termination. For discontinued subjects who will not revisit the clinic, the site will perform scheduled phone calls for the collection and source documentation for safety information (AEs, concomitant medication, and date of last dose
- Fitzpatrick skin type assessment should be done once before randomization.

#### 3.2.1 Screening Phase

Screening assessments will be performed up to 42 days prior to Day 1 of the double-blind treatment period. All screening evaluations must be completed and reviewed to confirm that potential subjects meet all eligibility criteria.

#### 3.2.2 Rescreening

If a subject has not met all eligibility criteria at the end of the Screening period, the subject will be registered as a screen fail. Screen fail subjects may be eligible for rescreening 1-time following consultation with the Sponsor and Medical Monitor.

Rescreened subjects must first be registered as screen failures and subsequently registered as rescreens. Once the subject is registered as rescreened, a new screening window will begin. The rescreened subject will be reassigned a new unique Subject Identifier and the previous Subject Identifier will be noted. If the rescreening period begins more than 30 days after the original signing of the ICF, all screening procedures, including ICF, must be repeated.

If the subject does not meet eligibility criteria for laboratory tests, the subject may undergo repeat laboratory tests up to 2 additional times during the 6-week Screening period. Repeat of laboratory tests is not considered rescreening.

#### 3.3 Sample Size and Power Considerations

For the primary estimand, the sample size of 159 is expected to provide adequate power for the comparisons between MT-7117 and placebo for change from baseline in the average daily sunlight exposure time (minutes) to first prodromal symptom associated with sunlight exposure between 1 hour post sunrise and 1 hour pre-sunset at Week 26 based on the MT-7117-A01 study. The calculation of sample size assumes a 2-sided alpha level of 0.05 and a 20% dropout rate up to Week 26. The sample size of 42 completers per treatment group will provide 91% and 79% power to detect an effect size of 0.72 and 0.66 in the average daily time (minutes) to first prodromal symptom associated with sunlight exposure between 1 hour post sunrise and 1 hour pre-sunset at Week 26 (ie, an absolute treatment difference of 57 mins between MT-7117 vs placebo, 52 mins between MT-7117 vs placebo, and a standard deviation [SD] of 79.3 mins). The sample size of 42 completers was calculated by SAS simulation using the fixed sequence testing procedure in order to confirm the power affected by multiplicity adjustment in treatment comparison for primary endpoint. Taking into account for a 20% dropout rate up to Week 26, total sample size of 159 was calculated.

Due to the rapid enrollment rate in the last few months of the enrollment period after COVID-


19 restrictions were lifted in many countries, a total of 184 subjects were enrolled.

#### 4 PLANNED ANALYSIS

The following analyses related to the objectives will be done twice in this study, Primary Week 26 Analysis and Final Analysis.

#### 4.1 Primary Week 26 Analysis

Primary Week 26 analysis will take place when the last subject completes Week 26 visit or follow-up period after DBT early termination and includes all subject data collected until then except for ongoing DBE or Follow up data. The available data in this analysis is as below;

| Subject<br>Type | Subject's Status on the date of LPLV for DBT | | | Primary Week 26 Analysis | | | |
|---|---|---|---|---|---|---|---|
| | DBT Period (26 weeks) | DBE Period<br>(26 weeks) | Follow up<br>(6 weeks) | DBT<br>data | DBE<br>data | Follow-<br>up data | FU Type |
| Α | Completed | Completed or Discontinued | Completed | X | х | X | DBE |
| В | Completed | Completed or Discontinued | No data | X | X | | |
| C | Completed or Discontinued | No data | Completed | X | | X | DBT |
| D | Completed or Discontinued | Ongoing in eith<br>/ No | ner DBE or FU<br>data | X | | | |

Note: X is "Included" in Primary W26 Analysis

After Week 26 database lock, the primary efficacy analysis will be conducted. No alpha adjustment for final analysis is needed, as this Week 26 efficacy analysis will be the primary efficacy analysis. The results will not be disclosed to any site-facing personnel or to any personnel directly involved with the conduct of the study. This detail was described in "MT-7117-G01 Blinding and Unblinding Plan Version 1.2 final.docx".

#### 4.2 Final Analysis

Final Analysis will take place when the patient data collected up to the time the last subject completes the last visit of Week 58 visit, unless last subject is lost to follow-up. This analysis will include all of the data in Primary Week 26 Analysis, and may include updated to partial or imcomplete data previously included in Primary Week 26 Analysis.

#### 5 ANALYSIS POPULATIONS

#### 5.1 Randomized (RAND) Population

The randomized (RAND) population includes all randomized subjects.

#### 5.2 Safety (SAF) Population

For the DBT data analysis

Safety Population 1 (SAF1) includes all randomized subjects who received at least 1 dose of study medication after randomization.

For the DBE data analysis

Safety Population 2 (SAF2) includes all randomized subjects who received at least 1 dose of study medication during DBE period.

The safety populations will be used for all safety analyses. The subject actual treatment received will be used for safety analyses. For subjects who took more than one treatment, the highest dose level will be used for safety analyses.

#### 5.3 Intent-to-treat (ITT) population

For the DBT data analysis

Intent-to-treat population 1 (ITT1) includes all randomized subjects who received at least 1 dose of study medication with baseline and post-randomization sunlight exposure diary assessment.

For the DBE data analysis

Intent-to-treat population 2 (ITT2) includes all randomized subjects who received at least 1 dose of study medication with baseline and post-randomization sunlight exposure diary assessment <u>during DBE period</u>.

The ITT populations will be used for all efficacy analyses. The subject randomized treatment will be used for efficacy analyses.

#### 5.4 Pharmacokinetic (PK) population

Pharmacokinetic (PK) population for the primary Week 26 analysis includes all randomized subjects who receive at least 1 dose of MT-7117 and who have at least 1 postdose value for plasma concentration at time point to be included in the PK analysis without important protocol deviations which may affect the PK of MT-7117.

PK population for the final analysis includes all randomized subjects who receive at least 1 dose of MT-7117 and who have at least 1 postdose value for plasma concentration at time point to be included in the PK analysis without important protocol deviations which may affect the PK of MT-7117.

#### 6 STATISTICAL CONSIDERATIONS

#### 6.1 Descriptive Statistics

Continuous data will be summarized descriptively using the number in the analysis set (N), the number of observations (n), mean, standard deviation (SD), median, minimum and maximum. Categorical data will be summarized using frequency counts and percentages. The denominator for the percentages will be the total number of subjects in the treatment group and analysis population being presented, unless otherwise specified (e.g. on some occasions, percentages may be calculated out of the total number of subjects with available data at a particular visit and/or time point).

Unless otherwise specified, all data will be summarized by analysis visits and treatment group.

#### 6.2 Statistical Tests

Unless otherwise specified, all formal statistical tests of treatment effects will be done at two-sided significance level of 0.05. Point estimates will be accompanied with two-sided 95% CIs where applicable.

#### 6.3 Stratification registration errors



patients. Therefore, it is planned to summarize the status of randomization factor registration error in the section of stratification registration errors and perform the sensitivity analysis for the primary efficacy endpoint to investigate the impact by the errors for study outcome.

#### 6.4 Dosing suspension

One case (Subject ID: with 3 serious adverse events (SAEs; cholestasis, ALT increased, and AST increased) was reported in this study. The SAE of cholestasis led to drug discontinuation and was fatal in this subject with a significant history of hepatic disease (i.e., cholestasis). The Investigator assessed the fatal SAE as probably related to study drug and the Sponsor assessed the fatal SAE as unlikely/unrelated to study drug. The principal investigator at the site 108 contacted their IRB in early July 2021 with their SAE assessment. As a result, the central IRB in the US requested a suspension of dosing for this study to MTDA and PI for US sites on July 14th 2021. Subsequently, the IRB released the dosing suspension on July 20th 2021 and allowed the US sites to resume dosing on the 21st July 2021. This dosing suspension gave some impact on dosing status for all ongoing subjects at every US site. Therefore, it is planned to summarize the status of dosing suspension in the section of treatment duration and compliance and perform the subgroup analysis of study drug compliance for the primary efficacy endpoint to investigate the impact by this drug suspension for the study outcome.

#### 7 DATA CONVENTIONS

Prior to the database lock, a blinded data review meeting for Primary Week 26 Analysis and a data review meeting for Final Analysis were conducted. Protocol deviations, protocol defined analysis populations and analysis visits were confirmed during these meetings (Blind Data Review Meeting minutes for Primary Week 26 analysis and Data Review Meeting minutes for Final analysis).

#### 7.1 Treatment Group Definitions and The Corresponding Analyzed Period Data

Two treatment group definitions for DBT data analysis and for DBE data analysis will be used as follows:

#### For DBT period data analysis

All DBT period data in all Subject type and Follow up period data in Subject type A, B, C and D in Section 4.1 will be analyzed with the below definition.

| Treatment Group | Definition 4 2 22 | |
|-----------------|----------------------|---------------------|
| MT-7117 | Allocated to MT-7117 | group in DBT period |
| MT-7117 | Allocated to MT-7117 | group in DBT period |

| Tresimitati/Group | Definition and the second |
|-------------------|------------------------------------------|
| Placebo | Allocated to Placebo group in DBT period |

#### For DBE period data analysis

All DBE period data and all Follow up period data in Subject Type A and B in Section 4.1 will be analyzed with the below definition.

| Treatment Group. | se Definition as a second | |
|-------------------------|---------------------------|----------------------|
| MT-7117 | Allocated to MT-7117 | group in DBT period |
| | and Enrolled in DBE peri- | od. |
| MT-7117 | Allocated to MT-7117 | group in DBT period |
| | and Enrolled in DBE peri- | od. |
| MT-7117 | Allocated to Placebo grou | |
| (switched from Placebo) | switched to MT-7117 | group in DBE period. |
| MT-7117 | Allocated to Placebo grou | p in DBT period and |
| (switched from Placebo) | switched to MT-7117 | group in DBE period. |

#### 7.2 Analysis Variable Definitions

#### 7.2.1 Study Subjects

#### 7.2.1.1 Protocol Deviation

Protocol deviations was be documented, reviewed, and determined in the blinded data review meeting for Primary Week 26 Analysis. The major protocol deviations that potentially influence the evaluation of the primary endpoint were selected in this meeting (Blind Data Review Meeting minutes for Primary Week 26 analysis).

#### 7.2.1.2 Demographic and Other Baseline Characteristics

#### (1) BMI

BMI will be recalculated using the formula below and reported to 1dp. BMI  $(kg/m^2)$  = weight at screening (kg) / {height at screening (m)}<sup>2</sup>.

#### (2) Disease Duration

Disease Duration (days) = the date of informed consent – the date of diagnosis+ 1. Disease Duration (years) = Disease Duration (days) / 365.25.

#### 7.2.1.3 Medical History

Medical history will be coded according to the MedDRA version 23.1.

#### 7.2.1.4 Prior or Concomitant Medication

Medications will be coded according to the WHO Drug Dictionary (WHO-DD) B3 MAR 2019 version.

#### (1) Prior Medication

Prior medications are defined as any medication taken within 1 month before the start date of study drug.

Any prior medication, including prescription and over-the-counter medications, taken within 1 month before Screening will be recorded on the eCRF. Information recorded will include: name of medication, dose, duration of and reason for use. It should be noted if subjects have ever used afamelanotide.

#### (2) Concomitant Medication

Concomitant medication is defined as any medication, other than study medication, which is taken during the study after the start date of study drug, including prescription, over-the-counter medications, herbals, dietary supplements, and recreational drugs. All concomitant medications taken while the subject is participating in the study will be recorded. Concomitant medication will be given only if deemed necessary by the Investigator or the subject's personal physician.

#### Rules to determine prior medications and concomitant medications:

Medications with a stop date before the first date of study drug dosing will be considered prior medications. Medications with start date or stop date on or after the first date of study drug dosing or ongoing at study will be considered concomitant medications.

#### Rule to determine concomitant medication for pain:

If indication in the eCRF for the concomitant medications includes "Pain" or "pain", the drug was regarded as comitant use for pain.

#### 7.2.1.5 Treatment Duration and Compliance

#### (1) Treatment Duration

For DBT period, treatment duration (days) = end of treatment date in DBT period – first treatment date + 1

For DBE period, treatment duration (days) = end of treatment date in DBE period - first treatment date in DBE period + 1

The time period of treatment duration is as below;

- $1 \le \le 29 \text{ (days)}$
- 29 < = < 85 (days)
- 85 < = < 183 (days)
- >183 (days)

For subjects lost to follow up, the treatment end date is taken to be the date of their last visit in the treatment periods. Interruptions and dose changes are not taken into account for treatment duration.

#### (2) Treatment Compliance

Treatment compliance will be calculated using the formula below and reported to 1dp by treatment periods. Interruptions and dose changes are not taken into account for treatment duration.

Treatment duration(days) – number of days subject miss the medication

Treatment duration (days) × 100%

#### 7.2.2 Efficacy assessments

#### 7.2.2.1 The Sunrise and Sunset Time to Use

The primary and some secondary efficacy endpoints are derived from the diary data. The sunlight exposure time between 1 hour post sunrise and 1 hour pre-sunset will be used. For the subjects exposed to sunlight, the sunrise and sunset times will be calculated for the corresponding country or geographical area. If the subjects exposed themselves while based in the US, the sunrise and sunset times for the corresponding US state, federal district, islands, or territory will be used.

To calculate sunrise and sunset times anywhere in the world, we will use the algorithms published by the National Oceanic and Atmospheric Administration (https://www.esrl.noaa.gov/gmd/grad/solcalc/calcdetails.htm).

During the ongoing study, the subjects' geographical locations for sunlight exposure will be reviewed from time to time. The sunrise and sunset time for the US locations, other countries, cities, and geographical areas will be added into SDTM as needed. The last time new sunrise and sunset time will be added is 5 weeks before the last subject last visit in the study. In the event that a subject had sun exposure while being in the location for which no sunrise and sunset time is readily available, the time 6:00 and 18:00 will be used as sunrise and sunset time. This is a close approximation of the average sunrise and sunset time for the current accumulated study data in the US.

#### 7.2.2.2 Data Handling of eDiary records

- (1) If there is inconsistency between start date and end date of a record for sunlight exposure, the following handling rule will be adapted.
  - If recorded end date is later than start date, end datatime will be changed to 23:59 on the same day of the start date.
  - If recorded start date is later than end date/time, the record will not be used for analysis.
- (2) If there is inconsistency between start date/time and end date/time of a record for prodromal symptom or phototoxic reaction, the following handling rule will be adapted.
  - If recorded end date/time is later than start date/time, keep as it is.
  - If recorded start date/time is later than end date/time, the record will not be used for calculation each time duration but used for counting the number of each event or summarizing the intensity of each event.
- (3) How to handle missing data for prodromal symptom and phototoxic reaction start/end time:

For prodromal symptom and phototoxic reaction start/end date missing, complete with the following handling rule after sorting by subject, day, and the linked sunlight exposure start time.

For the end time of prodromal symptom and phototoxic reaction missing, the earliest datetime of following three datetime after the linked sunlight exposure end time will be used as the end datetime.

- 1. Start datetime of next sunlight exposure record
- 2. Start/end datetime of next prodrome symptom or phototoxic reaction record
- 3. 23:59 of the day of linked sunlight exposure record

For the start time of prodromal symptom and phototoxic reaction missing, the latest datetime of following three datetime will be used as the start datetime.

- 1. End datetime of prior sunlight exposure record.
- 2. Start/end datetime of prior prodrome symptom or phototoxic reaction record
- 3. 0:00 of the day of linked sunlight exposure record

For the start/end time of prodromal symptom and phototoxic reaction missing without a linked sunlight exposure record, complement with the same rules as above after sorting by subject, the entry date time.

- (4) How to handle overlapping of eDiary start/end time:
  - For sunlight exposure records, complete with the following handling rule after sorting by subject, day, and the linked sunlight exposure start time to remove the overlapping among records by subjects and day.
  - 1. Compare the record's end time with next record's start time.

2. Combine them into one record and use the latest end time if end time is after the next start time.

#### 7.2.2.3 Derivation Rule for Efficacy Endpoints from eDiary records

## 7.2.2.3.1. The average daily sunlight exposure time (minutes) to first prodromal symptom associated with sunlight exposure

The following is the procedure to calculate the average daily time to first prodromal symptom associated with exposure to sunlight after removing overlapping among records. The analysis windows are defined in the Table 2 Analysis Visit Window for diary data.

- 1. If the sunlight exposure time is beyond the interval (from 1 hour post sunrise to 1 hour pre-sunset), then this time is excluded by comparing the sunrise/sunset time.
- 2. A diary day is qualified if the subject had non-zero duration of sunlight exposure in the day.
- 3. The time to first prodromal symptom associated with exposure to sunlight in a day is calculated. It is the sum of the sunlight exposure time before occurring the first prodromal symptom or phototoxic reaction associated with sunlight exposure (which means to occur after 1st sunlight exposure in a day) in the day. If a subject had sunlight exposure but no prodromal symptom in a day, the sum of the sunlight exposure time for the day is used as the sunlight exposure time to the first prodromal symptom.
- 4. The average daily sunlight exposure time to the first prodromal symptom at a time point (Baseline, Week 2, 4, 6, 8, 10, 12, 14, 16, ..., 24, 26, 39, 52 and Follow-up for each period) is the average of the sunlight exposure time to the first prodromal symptom of qualified days in the corresponding 14 day window. At least 1 day diary data is required for each 14 day window to be qualified for this calculation.
- 5. The minute is used as the unit for calculation of the duration. The duration will not be rounded. However, in data presentation for listings, the duration will be rounded to integer. For tables, the duration will be rounded to integer for minimum and maximum and to one decimal place for mean, SD, median, and confidence intervals.

# 7.2.2.3.2. The average daily mean intensity on an 11-point Likert scale of the subject's prodromal symptoms

The following is the procedure to calculate the average daily mean intensity on an 11-point Likert scale of the subject's sunlight-induced (equal to associated with sunlight exposure)

prodromal symptoms . The analysis windows are defined in the Table 2 Analysis Visit Window for diary data.

- 1. A day without any prodromal symptoms is not qualified.
- 2. The mean intensity on an 11-point Likert scale of the subject's prodromal symptoms in a day is calculated. It is the average of all the intensity on an 11-point Likert scale of the subject's sunlight-induced prodromal symptoms in the day. The average daily mean intensity on an 11-point Likert scale of the subject's prodromal symptoms at a time point (Baseline, Week 2, 4, 6, 8, 10, 12, 14, 16, ..., 24, 26, 39, 52 and Follow-up for each period) is the average of the daily mean intensity of qualified days in the corresponding 14 day window. At least 1 day diary data is required for each 14 day window to be qualified for this calculation.

The following endpoint is derived when applying the similar rule as above.

- The average daily mean intensity of the subject's phototoxic reactions (associated with sun exposure) on an 11-point Likert scale

# 7.2.2.3.3. The average daily duration of sunlight exposure regardless of time of day without prodromal symptoms

The following is the procedure to calculate the average daily mean duration of sunlight exposure regardless of time of day without prodromal symptoms. The analysis windows are defined in the Table 2

- 1. Step 1 in section 7.2.2.3.1 will not be applied.
- 2. A diary day is qualified if the subject had non-zero duration of sunlight exposure in the day.
- 3. The duration of sunlight exposure without prodromal symptoms in a day is calculated. It is the sum of the duration of sunlight exposure time deducting the prodromal symptom or phototoxic reaction presenting time covered in each period.
- 4. Step 4 to 5 in section 7.2.2.3.1 will be applied.

# 7.2.2.3.4. Total number of sunlight-induced pain events defined as prodromal symptoms (burning, tingling, itching, or stinging) with pain rating of 1-10 on the Likert scale

The following is the procedure to calculate this endpoint.

- 1. If a subject had sunlight exposure with any prodromal symptom with pain rating of 1-10 on the Likert scale in a day, the sum of the number of events for the day is used as the number of sunlight-induced pain events in the day.
- 2. The sum of the number of the above events in each day during the 26-week DBT or DBE period (from Baseline date to Week 26 or from Week 26 to Week 52) is calculated as this endpoint.

The following endpoint is derived when applying the similar rule as above.

- Total number of sunlight-induced non-prodrome, phototoxic reactions
- Total number of sunlight-induced pain events defined as phototoxic events

# 7.2.2.3.5. Total time (hours) in duration of sunlight exposure between 1 hour post sunrise and 1 hour pre-sunset without prodromal symptoms.

The following is the procedure to calculate this endpoint.

- 1. Step 1 in section 7.2.2.3.1 will be applied.
- 2. The duration of sunlight exposure without prodromal symptoms and without phototoxic reactions in a day is calculated.
- 3. The sum of the above duration in each day during the 26-week DBT or DBE period (from Baseline date to Week 26 or from Week 26 to Week 52) is calculated as this endpoint.

The following endpoint is derived when applying the similar rule as above. Total time (hours) in duration of sunlight exposure between 1 hour post sunrise and 1 hour pre-sunset without prodromal symptom with the severity of greater than 0 on 11-point Likert scale and without phototoxic reactions (pain-free time hours)

The following endpoint is derived as pain-free days when applying the similar rule as above.

- Total number of days subject is exposed to sunlight for any duration between 1 hour postsunrise and 1 hour pre-sunset without prodromal symptoms
- Total number of days subject is exposed to sunlight for any duration between 1 hour postsunrise and 1 hour pre-sunset without prodromal symptom with the severity of greater than 0 on 11-point Likert scale and without phototoxic reactions (pain-free days)

#### 7.2.2.4 PGIC

The following score will be assigned and used for each outcome.

1: Very Much Improved

- 2: Much Improved
- 3: Minimally Improved
- 4: No Change
- 5: Minimally Worse
- 6: Much Worse
- 7: Very Much Worse

#### 7.2.2.5 PGIS

The following score will be assigned and used for each outcome.

- 1: None
- 2: Mild
- 3: Moderate
- 4: Severe
- 5: Very Severe

#### 7.2.2.6 PROMIS-57

Raw score for each PROMIS domain will be calculated as follows:

- Physical function raw score= total of Question 1 (PRO001) Question 8 (PRO008)
- Anxiety raw score = 48 (=6x8) total of [Question 9 (PRO009) Question 16 (PRO016)]
- Depression raw score = 48 (=6x8) total of [Question 17 (PRO017) Question 24 (PRO024)]
- Fatigue raw score = 48 (=6x8) total of [Question 25 (PRO025) Question 32 (PRO032)]
- Sleep Disturbance raw score = 48(=6x8) total of [Question 33 (PRO033) Question 40 (PRO040)]
- Ability to Paricipate in Social Roles and Activities raw score = total of Question 41 (PRO041) Question 48 (PRO048)
- Pain Interference = Pain Intensity = 0 (No pain) to 10 (Worst pain imaginable) numeric rating scale (Categorical)

Total raw score for PROMIS all domain will be calculated as follows:

• The mean of physical function raw score, anxiety raw score, depression raw score, fatigue raw score, sleep disturbance raw score, ability to participate raw score, pain interference rawscore.

If there is missing score data in an domain or total, the corresponding domain or total score will be missing.

#### 7.2.3 Safety Assessments

#### 7.2.3.1 Adverse Events

Adverse events will be coded according to the MedDRA version 23.1.

(1) Treatment Emergent Adverse Events/ Treatment Emergent Serious Adverse Events (TEAEs/TESAEs)

AEs will be classified as 'treatment-emergent' if they arise following the first administration of study medication in the treatment period (after randomization) or if a pre-dose AE increases in severity following dosing in the treatment period (after randomization).

#### Rule to determine TEAE using onset date of AEs:

An AE is classified as treatment emergent if it newly occurred on or after the first dose of study drug. According to this data handling, for the severity part in the above TEAE definition, the AE with upgraded severity and with the new onset date during the treatment period will be automatically included as TEAE.

#### (2) Adverse Event Related to Study Drug

A TEAE is considered "adverse event related to study drug" if it has been assessed as having a "reasonable possibility" in relationship to the study drug.

#### (3) Duration of Adverse Events

Duration of Adverse Events (days) = AE stop date – AE start date + 1.

#### (4) Time to AE onset

For DBT period, time to AE onset (days) = AE start date – the first treatment date in DBT period + 1.

For DBE period, time to AE onset (days) = AE start date – the first treatment date in DBE period + 1.

#### 7.2.3.2 Physical examiniation

If "Abnormal, Unchanged from previous assessment" is selected and there is no available data of "Clinically Significant" or "Not Clinically Significant" in the previous assessment, the analysis value will be regarded as "Abnormal, Clinically Significant".

#### 7.2.3.3 Laboratory Tests

(1) Criteria for pre-defined limit

#### Liver function:

- ALT  $\geq$  10 × ULN
- $8 \times ULN \le ALT \le 10 \times ULN$
- 5×ULN <= ALT < 8×ULN
- $3\times ULN \le ALT < 5\times ULN$
- 1×ULN <= ALT < 3×ULN

The above same criteria will be applied to AST.

- Total Bilirubin >= 2×ULN
- 1×ULN <= Total Bilirubin <2×ULN

#### 7.2.3.4 12-Lead ECG

(1) Criteria for pre-defined limit

#### 12-lead ECG:

- Baseline QTc <450 msec and >500 msec at any post baseline
- Baseline QTc <450 msec and 500 msec  $\geq$  QTc >480 msec at any post baseline
- Baseline QTc <450 msec and 480 msec  $\geq$  QTc >450 msec at any post baseline
- Increase from baseline in QTc > 30 msec, 60msec at any post baseline

The above same criteria will be applied to QTcF and QTcB.

#### 7.2.4 Data Handling of PK data and melanin density data

The PK data and melanin density (MD) data handling will be confirmed during blinded data review (BDR). PK data and MD data that are considered "invalid" will be flagged in the listing and will be excluded from the calculation of summary statistics. Due to the nature of PK data and MD data, some issues may only be discovered after PK data and MD data are unblinded. Should new issues be identified post unblinding, and new data handling rules would have to be applied, a separate PK data and MD data handling document will be produced to provide detailed rationale and decision making. If there is clear evidence that PK sample handling errors, MD handling errors, or other factors are identified after data unblinding and these errors have led to unexpected erroneous data, then these erroneous data will be regarded as "invalid", full explanations will be given in the PK data and MD data handling document.

#### 7.3 Analysis Visit Definitions

#### (1) eDiary data excluding in-clinic sunlight exposure test

The subjects will, in their diaries, record the sunlight exposure periods (start/end time), prodromal symptom periods, and pain periods. The subjects' sunlight exposure start and end times will be compared with their state capital cities sunrise and sunset times.

The analysis windows are defined in the table below. The nominal day for each week relative to the first dose day will be used. Day 1 is the first dose day.

Table 2 Analysis Visit Window for diary data

| Analysis Visit | Nominal day | Analysis Visit Window for DBT analysis |
|---|---|---|
| Baseline* | Day 1 | Day -14 to -1 |
| Week 2 | Day 15 | Day 1 to 14 |
| Week 4 | Day 29 | Day 15 to 28 |
| Week 6 | Day 43 | Day 29 to 42 |
| Week 8 | Day 57 | Day 43 to 56 |
| Week 10 | Day 71 | Day 57 to 70 |
| Week 12 | Day 85 | Day 71 to 84 |
| Week 14 | Day 99 | Day 85 to 98 |
| Week 16 | Day 113 | Day 99 to 112 |
| Week 18 | Day 127 | Day 113 to 126 |
| Week 20 | Day 141 | Day 127 to 140 |
| Week 22 | Day 155 | Day 141 to 154 |
| Week 24 | Day 169 | Day 155 to 168 |
| Week 26 (DBT EOT) | Day 183 | Day 169 to 182 |
| Week 26 (DBE | Day 183 | Day 169 to 182 |
| Baseline) | | |
| Week 28 | Day 197 | Day 183 to 196 |
| Week 32 | Day 225 | Day 211 to 224 |
| Week 39 | Day 274 | Day 260 to 273 |
| Week 52 (DBE EOT) | Day 365 | Day 351 to 364 |
| EOT for DBT | Day 182 or discontinued during DBT | 14 days before EOT for DBT |
| EOT for DBE | Day 365 or discontinued during DBE | 14 days before EOT for DBE |
| Follow-up until Week | 6 weeks after EOT for | the latest 1 to 14 days before |
| 32 (DBT EOS) | DBT | Follow-up date not |
| | | overlapping with treatment |
| | | duration in DBT period |
| Follow-up until Week | 6 weeks after EOT for | the latest 1 to 14 days before |
| 58 (DBE EOS) | DBE | Follow-up date not |
| | | overlapping with treatement |
| | | duration in DBE period |
| During 26 weeks<br>(DBT) | 1 to 182 | Day 1 to EOT for DBT period |
|--------------------------|------------|------------------------------------|
| During 26 weeks<br>(DBE) | 183 to 364 | DBE Baseline to EOT for DBE period |

<sup>\*</sup> If subjects have at least 1 day between Day -1 and Day -14, the baseline value will be calculated from the data between Day -1 and Day -14. If subjects have no data of sunlight exposure between Day -1 and Day -14, then the Analysis Visit window will be expanded to Day -28 and the baseline value will be calculated from the data between Day -1 and Day -28.

# (2) Non-diary data including in-clinic sunlight exposure test

Table 3 Analysis Visit Window for non-diary efficacy data

| Analysis Visit | Nominal day | Analysis Visit<br>Window |
|---|---|---|
| Baseline | First dose day | NA |
| Week 4 | Day 29 | Day 16 to 64 |
| Week 12 | Day 85 | Day 72 to 119 |
| Week 26 (DBT EOT) | Day 183 | Day 134 to 202 |
| Week 26 (DBE Baseline) | Day 183 | Day 134 to 202 |
| Week 39 | Day 274 | Day 250 to 320 |
| Week 52 (DBE EOT) | Day 365 | Day 321 to 396 |
| Follow-up until Week 32 (DBT EOS) | 6 weeks after EOT for DBT | NA |
| Follow-up until Week 58 (DBE EOS) | 6 weeks after EOT for DBE | NA |

## (3) Safety data

Table 4 Analysis Visit Window for safety data

| Analysis Visit | Nominal day | Analysis Visit<br>Window |
|------------------------|-----------------|--------------------------|
| Screening* | Day -42* | - |
| Baseline* | First dose day* | NA* |
| Week 2 | Day 15 | Day 2 to 22 |
| Week 4 | Day 29 | Day 23 to 42 |
| Week 8 | Day 57 | Day 43 to 71 |
| Week 12 | Day 85 | Day 72 to 119 |
| Week 16 | Day 113 | - |
| (Only for Norway site) | | |
| Week 18(Only for Japan | Day 127 | - |
| and Canada site) | | |
| Week 20 | Day 141 | - |
| (Only for Norway site) | | |
| Week 26 (DBT EOT) | Day 183 | Day 134 to 190 |

| Week 26 (DBE Baseline) | Day 183 | Day 134 to 190 |
|---|---|---|
| Week 28 | Day 197 | Day 191 to 211 |
| Week 30 | Day 211 | |
| (Only for Germany site) | | - |
| Week 32 | Day 225 | Day 212 to 249 |
| Week 36 | Day 253 | |
| (Only for Norway, | | - |
| Germany and Canada site) | | |
| Week 39 | Day 274 | Day 250 to 320 |
| Week 43 | Day 302 | - |
| (Only for Norway site) | | |
| Week 47 | Day 330 | - |
| (Only for Norway site) | | |
| Week 52 (DBE EOT) | Day 365 | Day 321 to 396 |
| EOT for DBT | Day 182 or discontinued during DBT | The latest visit during |
| (LOCF) | | DBT period |
| EOT for DBE | Day 365 or discontinued during DBE | The latest visit during |
| (LOCF) | | DBE period |
| Follow-up until Week 32 | 6 weeks after EOT for DBT | NA |
| (DBT EOS) | | INC |
| Follow-up until Week 58 (DBE EOS) | 6 weeks after EOT for DBE | NA |
| (DDE EUS) | | |

<sup>\*</sup> For liver function markers (ALT, AST, GGT, ALP, direct and total bilirubin), the mean value of two numerical values at screening visit and at randomization visit (the first dose day) will be treated as a baseline value.

The date of the first dose of study drug is defined as Day 1.

Unless otherwise specified, baseline will be the last observed value of the parameter of interest prior to the first intake of study drug (for DBT) or will be the available value of parameter of Week 26 (for DBE).

For other visits, if there are multiple data in a window, the closest data to nominal day will be used. If the distance to the nominal day is the same, the data of later date will be used.

According to country specific protocol for Japan, Norway, Germany and Canada, liver function markers (ALT, AST, GGT, ALP, direct and total bilirubin) will be measured at each country specific visit in each country.

### 7.4 Data Handling Convention for Missing Data

For missing of the onset time of the first prodromal symptom in in-clinic sunlight exposure test, impute from the formula of "end test time - start test time" as sensoring time.

For the purpose of determining TEAE and AE duration, if the AE start date is incomplete, it will be imputed as follows:

- If the start date is completely missing, the start date will be equal to the date of the first dose date of study treatment. However, if the stop date is not missing and is before the date of the first dose of study treatment, then the stop date will be used instead and the AE will not be considered as TEAE.
- If the start day is missing, but the month and year are not missing and are equal to the month and year of the first study dose, then this event will be considered as TEAE.
- If the start day and month are missing, then the first day of the first month (January) will be used.

If an AE stop date is incomplete, it will be imputed as follows for the purpose of determining AE duration:

- If the AE stop date is completely missing, then the stop date will be equal to the subject's last observed date.
- If the Stop day is missing, but the month and year are not missing and are equal to the month and year of the last observed date, then stop date will be equal to last observed date.
- If the start day and month are missing, then the first day of the first month (January) will be used.

For the purpose of determining prior and concomitant use, if the medication start date is incomplete, then it will be imputed as follows:

- If the start date is completely missing, the start date will be equal to the first dose date. However, if the stop date is not missing and is before the first dose date, then the stop date will be used instead.
- If the start day is missing, the first day of the month will be used.
- If the start day and month are missing, then the first day of the first month (January) will be used.

If the medication stop date is partial, then it will be imputed as follows for the purpose of determining prior and concomitant use:

- If the stop date is completely missing and the medication is not ongoing, the stop date will be equal to the last dose date or date of completion/withdrawal, whichever is the latest.
- If the stop day is missing, the last day of the month will be used.
- If the stop day and month are missing, then the last day of the last month (December) will be used.

#### 8 STATISTICAL METHODOLOGY

Listings will be presented in treatment, subject, visit (where applicable), and date (where applicable) order.

### 8.1 Study Subjects

#### 8.1.1 Subject Disposition

Subject disposition will be summarized on the RAND population.

The number of subjects who completed all treatment period (DBT and DBE), prematurely discontinued either DBT period or DBE period, completed DBT period, DBE period, and the safety follow-up period with the reasons for discontinuation in each period will be summarized. In addition, the number and percentage of the subjects that received placebo treatment in MT-7117-A01 study will be summarized.

The number of subjects who enter screening will be summarized, and the percentage of these subjects who fail to meet entry criteria will be reported for total subjects. Screen failures will be summarized in total and by each reason for screen failure.

#### 8.1.2 Analysis Populations

Analysis populations will be summarized on the RAND population. Analysis populations will be listed on the RAND population.

#### 8.1.3 Protocol Deviations

Protocol deviations including major deviations specified in the blinded blinded data review meeting will be listed on the RAND population.

#### 8.1.4 Stratification Registration Errors

In addition, the number of subjects with unmatched stratification registration will be summarized by comparing between IWRS strata data and actual strata from e-Diary data derivation and between IWRS strata data and vendor report strata on the RAND population.

#### 8.1.5 Demographic and Other Baseline Characteristics

The following demographic and other baseline characteristics will be used.

| | Category | Descriptive |
|---|---|---|
| Sex | Male, Female | |
| Age (years) | Adolescent(<18)<br>Adult(18 – 65, >65) | Yes |
| Height (cm) at screening visit | | Yes |
| Weight (kg) at screening visit | <45<br>>=45 | Yes |
| BMI (kg/m2) | | Yes |
| Race | White, Black or African American, Asian(Japanese), American Indian or Alaska Native, Native Hawaiian or Pacific Islander, Other | |
| Country | US, Australia, Canada,<br>Germany, Italy, Japan, Norway,<br>Spain, Sweden, United Kingdam<br>(from IWRS data) | |
| Region (Randomization stratification factor) | North America, Rest of world (Europe, Japan, Australia) (from IWRS data) | |
| Ethnicity | Hispanic or Latino,<br>Non-Hispanic or Latino | |
| EPP/XLP | EPP,<br>XLP | |
| Protoporphyrin (PPIX level) (mcg/dL) | | Yes |
| Disease duration (years) | | Yes |
| Baseline average daily time to<br>first prodromal symptom<br>(Randomization stratification<br>factor) | | |
| Actual baseline average daily time to first prodromal symptom | | Yes |
| Seasonality 1 | Randomized in Spring and Summer inclusive, Other | |

| | (Spring and Summer: between<br>September 1st to February 29 in<br>Australia<br>or<br>between March 1st and August<br>31th in the other countries) | |
|---|---|---|
| Seasonality 2 | Week 26 visit in Spring and Summer inclusive, Other (Spring and Summer: the date of Week 26 analysis visit is between September 1st and February 29th in Australia or the date of Week 26 analysis visit is between Mar 1st and August 31th in the other countries) | |
| Melanin density | | Yes |
| Fitzpatrick skin type | Ι, Π, ΙΠ, ΙV, V-VΙ | |

Demographic and other baseline characteristics will be summarized on the ITT1, ITT2, SAF1, and SAF2 populations. Demographic and other baseline characteristics will be summarized on the ITT1, ITT2, SAF1, and SAF2 populations by region (North America, Europe, Japan, Australia).

Demographic and other baseline characteristics will be listed on the RAND population.

#### 8.1.6 Medical History

| Medical history wi | Ill be summarized on | the SAF1 and the SAF2 population | ulations. In this summary |
|---|---|---|---|
| SOC is sorted by International order; then within SOC, PT is sorted by descending counts | | | |
| under MT-7117 | , MT-7117 | or Placebo (switched to | , switched to |
| ) column, th | en alphabetic order f | for PTs with the same count. I | Medical history will be |
| listed on the RANI | D population. | | |

#### **8.1.7** Prior or Concomitant Medications

The prior will be summarized in table separately by ATC level 2, preferred name and treatment group for the SAF1 and presented in data listing for the RAND population. The concomitant medications that were used based on the start date of use during each period of DBT and DBE will be summarized by ATC level 2, preferred name and treatment group for the SAF1 and SAF2 populations respectively and presented in data listing for the RAND population.

#### 8.1.8 Prohibited medication

The prohibited medications coded by the protocol Appendix 1 Table 18-1 will be summarized on the SAF1 and SAF2 populations and listed on the RAND population. The summary will be presented by ATC level 2 and preferred name and treatment.

#### 8.1.9 Treatment Duration and Compliance

Treatment duration will be summarized on the ITT1 and ITT2 populations.

Treatment duration and compliance will be listed on the RAND population. Study drug interruptions will be listed on the RAND population.

Compliance to Double-Blind study medication will be presented for the ITT1 and ITT2 population in table by treatment group. The range 80% <= compliance <= 120% will be used to define a subject being treatment compliant.

The number and percentage of subjects with no study drug suspension, any study drug suspension and permanent study drug discontinuation will be summarized by the DBT period on the ITT1 population and by the DBE period on the ITT2 population.

All study medication administration and accountability data will be listed by subject.

#### 8.1.10 Fitzpatrick skin scale test

The Fitzpatrick skin type will be summarized with number and percentage and the Fitzpatrick total score will be summarized by treatment group and analysis visit for the ITT1 and ITT2

populations.

### 8.1.11 Subject Questionnaire for Study Medication

Subject questionnaire for study medication will be summarized and listed.

### 8.2 Efficacy Assessments

All efficacy endpoints will be analysed under primary estimand unless otherwise stated. All data will be listed.

#### For DBT data analysis

All efficacy endpoints in Section 2.3.1, 2.3.2, and 2.3.3 will be summarized using descriptive statistics or using the number with percentage in the ITT1 population. All of the statitistical model analyses stated in the below sections will be done in the ITT1 only for DBT data analysis only.

#### 8.2.1 Primary Efficacy Endpoint

### **Primary Analysis**

For the ITT1 population, the primary estimand will be tested including retrieved dropout data (after treatment discontinuation), using treatment comparisons of interest in change from baseline in average daily time to first prodromal symptoms associated with exposure to sunlight between 1 hour post sunrise and 1 hour pre-sunset for the two MT-7117 doses ( and and compared with placebo at Week 26 (Visit 7).

To assess the treatment effect at Week 26, change from baseline in average daily time (minutes) to first prodromal symptom associated with exposure to sunlight between 1 hour post sunrise and 1 hour pre-sunset at Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, and 26 will be analyzed using mixed-effect model for repeated measures (MMRM). The model will include fixed categorical terms for treatment,

visit, and treatment by visit interaction together with continuous covariate terms for baseline average daily duration of sunlight exposure between 1 hour post sunrise and 1 hour pre-sunset to first prodromal symptom and baseline average daily duration of sunlight exposure between 1 hour post sunrise and 1 hour pre-sunset to first prodromal symptom by visit interaction. An unstructured (UN) correlation structure will be used to model the within-subject variance covariance errors. Should convergence of the model fail (due to the small numbers of

subjects in this study), the heterogeneous compound symmetry (CSH) and the heterogeneous Toeplitz structure (TOEPH), autoregressive [AR(1)] and compound symmetry (CS) correlation matrix will be used in that order instead of UN. The Kenward-Roger approximation will be used to estimate the denominator degrees of freedom. From the model described above, adjusted (least squares [LS]) means and standard errors will be produced by treatment group and visit. Difference in adjusted means at each visit (each MT-7117 dose vs. placebo) with standard errors, 95% CIs and associated p-values will also be produced. All available data from all subjects will be used in the primary analysis without any imputation.

#### Sensitivity Analysis

(1) Use of actual strata of baseline average daily sunlight exposure time to first prodromal symptom for randomization registration errors

In the above primary analysis model,

directly
derived from e-Diary raw dataset.

(2) Controlled multiple imputation method

The primary analysis model is using likelihood based approach to handle missing data under Missing At Random (MAR) missingness pattern in the primary estimand. In order to assess the robustness of the primary analysis also under Missing Not At Random (MNAR) pattern, a control group-based multiple imputation (MI) of the Pattern Mixture Model (PMM) method will be used. This model assumes MNAR for missing data mechanism in MT-7117 and and MAR for missing data mechanism in placbo on the ITT population.

- Step 1: This methodology will structure data based on missing data patterns. The PMM method will be based on a missingness pattern having a monotone structure, i.e. if among the observations over time one data value is missing, all other values after this missing value will also be missing. For patients with intermittent missing values, before performing MI based on the PMM, it will be necessary to create a monotone missingness pattern. Intermittent missing values will be imputed using the Markov Chain Monte Carlo (MCMC) methodology which assumes a multivariate normal distribution over all variables included in the imputation model. The MI procedure in SAS will be used for this purpose and this first MI step is planned to be repeated 100 times, creating different datasets with a monotone missing data structure. Seed value of 2022 will be used in the MI procedure. The imputation with the explanation variables of the baseline value and the post-baseline values is based on the MAR assumption, i.e. the missing data are assumed to follow the same model as the other patients. The minimum number

will be set as 0 because the imputed value for time to first prodromal symptom should be greater than or equal to 0.

| The following SAS code will be used to generate the monotone missing data pattern: |
|---|
| Step 2: After this, the remaining missing data will be imputed using a MI method for monotone missingness, with the assumption that the data on MT-7117 and and once daily groups are MNAR and the data on placebo group are MAR. Control group-based assumption will be used for the missing data. Thus, for each of the created dataset with a monotone missing data pattern in step 1, the MI procedure in SAS will be used to impute missing values based on a sequential procedure reflecting the monotone missing data pattern. The MNAR statement of the following (see SAS code) will be used to generate the imputation. |
| Patients with the first missing value occurring at Week 2 ("W2") will have their missing Week 2 value replaced by an imputed value from a regression model with and the |
| baseline value (BASE) as explanatory variables. In the next step, patients with their Week 4 ("W4") value missing will have their missing Week 4 value replaced by an imputed value from a regression model with baseline average daily first to prodromal symptoms and the Week 2 value as explanatory variables. Similar procedure will be used to replace the missing values at week 4, 6, 8 and 10 etc. |
| If the imputated value is less than 0 and then the valus will |
| be replaced with 0. |
| The following SAS code for the missing data imputation at Week 26 will be used to make the |
| imputation with the MNAR assumption: |

- Step 3: The imputed dataset (IMPUTED) generated with the approach described above do contain only non-missing values. MMRM model similar to that described for the primary analysis will thus be run on each of the 100 generated imputed datasets and the differences between the treatment groups at Week 26 will be estimated (and export to data 'ESTIMATES'). Finally, the MIANALYZE procedure in SAS will be applied to combine the results from these analyses to derive an overall estimate of the treatment differences at W26. In addition to the estimates, corresponding 95% confidence intervals and p-values will be calculated.



The following example SAS code will be used:

### (3) Non-parametric analysis

Non-parametric analysis will be performed in order to confirm the robustness for the above parametric model. The change from baseline in average daily time (minutes) to first prodromal symptom associated with exposure to sunlight between 1 hour post sunrise and 1 hour presunset at each visit (Weeks 2, 4,..., 24, and 26) from two treatments being compared will enter the corresponding analysis. The point estimates and two-sided 95% confidence intervals for the difference between the treatment groups will be obtained using the Hodges-Lehman estimator corresponding to Wilcoxon's rank sum test. The paired comparison between each MT-7117 arm with placebo will also be performed using this non-parametric analysis method. This nonparametric analysis will be performed with multiple imputation (MI) method in the following steps, assuming missing at random.

- MI Step 1: Intermittent missing values will be imputed using the Markov Chain Monte Carlo (MCMC) methodology which assumes a multivariate normal distribution over all variables included in the imputation model. The MI procedure in SAS will be used for this purpose and this first MI step is planned to be repeated 100 times, creating different datasets with a monotone missing data structure. Seed value of 2022 will be used in the MI procedure. The minimum number will be set as 0 because the imputed value for time to first prodromal symptom should be greater than or equal to 0.



- MI Step 3: The imputed datasets generated with the approach described above do contain only non-missing values and are used as input in the model for the sensitivity analysis for the primary efficacy endpoint. For the difference between the treatment groups with paired comparison

| Statistical Ar | alysis | Plan |
|----------------|--------|---------|
| Protocol No. | MT-7 | 117-G01 |

Mitsubishi Tanabe Pharma Development America

vs. Placebo and MT-7117 vs. Placebo) in Week 2, 4, ..., 24, and 26, the Hodges-Lehman estimator and asymptomtic standard error of this estimator will be calculated on each of the 100 generated imputed datasets, using the NPAR1WAY procedure in SAS. Finally, the MIANALYZE procedure in SAS will be applied to combine the results from these analyses to derive an overall estimate of the treatment differences at Week 2, 4, ..., 24, 26 according to the following code. In addition to the estimates, corresponding 95% confidence intervals and p-values will be calculated.

The following example SAS code will be used:



(3) LOCF imputation analysis

For this primary endpoint, ANCOVA with treatment group (trtp),

and the baseline value as the explanatory variables will be also performed. For missing data for the primary endpoint, LOCF approach assuming MNAR will be used to impute this missing data.

These three subjects data will be removed from the primary endpoint and the above primary analysis model will be performed.

### **Supportive Analysis**

The secondary estimand will use similar estimator as for the primary analysis. The ITT1 population with the primary efficacy data without retrieved dropout data (after treatment discontinuation) will be used for this analysis. Likelihood based model method under Missing at Random assumption will be performed using the same MMRM as specified for the primary analysis. The only primary endpoint will be also analyzed in the secondary estimand and the other efficacy endpoints will not be analyzed in this estimand.

## Multiplicity adjustment for treatment comparison on primary and secondary endpoints

The overall study-wise type I error will be 5%. Type I error will be globally strongly controlled by employing the fixed sequence approach, (i.e., each endpoint will be formally analyzed only in case the preceding endpoint will have a p-value less than or equal to 0.05).

To protect the study from type I error inflation, the lower ordered comparison will be interpreted inferentially only if a statistically significant treatment effect is detected in the higher ordered comparison (H1=>H2,..., H11=>H12). The following null hypothesis will be sequentially tested via the following order;

H1: There is no treatment difference between MT-7117 and and placebo in change from baseline in average daily time (minutes) to first prodromal symptom associated with exposure to sunlight between 1 hour post sunrise and 1 hour pre-sunset at Week 26.

H2: There is no treatment difference between MT-7117 and and placebo in change from

baseline in average daily time (minutes) to first prodromal symptom associated with exposure to sunlight between 1 hour post sunrise and 1 hour pre-sunset at Week 26.

H3: There is no treatment difference between MT-7117 and placebo in PGIC at Week 26.

H4: There is no treatment difference between MT-7117 and placebo in PGIC at Week 26.

H5: There is no treatment difference between MT-7117 and and placebo in total number of sunlight-induced pain events defined as prodromal symptoms (burning, tingling, itching, or stinging) with pain rating of 1-10 on the Likert scale during 26-week double-blind treatment period.

H6: There is no treatment difference between MT-7117 and and placebo in total number of sunlight-induced pain events defined as prodromal symptoms (burning, tingling, itching, or stinging) with pain rating of 1-10 on the Likert scale during 26-week double-blind treatment period.

H7: There is no treatment difference between MT-7117 and and placebo in change from baseline for total score in the domain of pain intensity in the PROMIS-57 at Week 26.

H8: There is no treatment difference between MT-7117 and and placebo in change from baseline for total score in the domain of pain intensity in the PROMIS-57 at Week 26.

H9: There is no treatment difference between MT-7117 and and placebo in the percentage of subjects who are responders at Week 26 based on average daily sunlight exposure time to first prodromal symptoms using the within-subject meaningful change of 66 minutes increase.

H10: There is no treatment difference between MT-7117 and and placebo in the percentage of subjects who are responders at Week 26 based on average daily sunlight exposure time to first prodromal symptoms using the within-subject meaningful change of 66 minutes increase.

H11: There is no treatment difference between MT-7117 and placebo in change from

baseline for total score in the domain of physical function in the PROMIS-57 at Week 26.

H12: There is no treatment difference between MT-7117 and placebo in change from baseline for total score in the domain of physical function in the PROMIS-57 at Week 26.

### **Subgroup Analysis**

The consistency of treatment effect on the primary endpoint across different subgroups will be explored based on the ITT1 population and the primary estimand for the following subgroups using the primary efficacy analysis.

- Gender (Male, Female)
- Age group (age <18, 18=< age)
- Tigo group (ago 110, 10 1 ago
- Ethnicity (Hispanic or Latino, Non-Hispanic or Latino, Others)
- Race (White, Black or African American, Asian(Japanese), Others)
- BMI (BMI  $\leq$ 30, BMI  $\geq$ 30 kg/m<sup>2</sup>)
- Seasonality1 (Randomized in Spring and Summer inclusive, Other)
- Seasonality2 (Week 26 visit in Spring and Summer inclusive, Other)
- Average melanin density at BL (>=Median, <Median)
- Fitzpatrick scale test category (I-II or III-VI)
- Protoporphyrin (>=Median, <Median)
- Porphyrin (>=Median, <Median)
- EPP vs XLP
- Study Drug Compliance by Week 26 (no study drug suspension, any study drug suspension or permanent study drug discontinuation)

# Bayesian analysis for adult and adolescent subgroups

Age group (age <18, 18=<age)

In order to estimate treatment effects for adult and adolescent for the primary endpoint, Bayesian subgroup hierarchical model and Commensurate prior model will be performed using both adolescent and adult subgroup data in order to get greater precision on treatment effect and address random high and random low data values due to small sample estimates. This means these analysis does not estimate treatment effect within adolescent subgroup in isolation of adult subgroup. Details of the model and the framework can be found in Appendix 1. The posterior means, SE and 95% Credible Interval(CrI) for the primary endpoint will be presented for each treatment group. The posterior mean, SE and 95% CrI will be obtained for the difference of each of the active MT-7117 treatment groups versus placebo. In addition, the probability that the difference in the primary endpoint versus placebo > 0 will be presented for MT-7117 and and present the primary endpoint versus placebo is at least greater than 95%, then this will be considered as "a statistically significant difference" for the active dose and the subgroup. If the posterior mean for the difference in the primary endpoint versus placebo will be greater than 0 in both adult and adolescent subgroups in the MT-7117 active dose, then this will be considered as "a positive trend" for the active dose among the subgroups.

### Funnel plot analysis

#### 8.2.2 Secondary Efficacy Endpoints

The secondary endpoint PGIC at Week 26 will be analyzed using the similar model as specified for the primary analysis (MMRM) replacing the average daily sunlight exposure time to first prodromal symptom baseline covariate with PGIS covariates at baseline visit.

The change from baseline for total score in each domain of physical function and pain intensity in the PROMIS-57 at Week 26 will be analyzed in the same way.

For the total number of sunlight-induced pain events defined as prodromal symptoms with pain rating of 1-10 on the Likert scale during the 26-week double-blind treatment period, the negative binomial regression model with log link will be used. The model will include treatment and the randomization stratification factors as fixed effect. The estimated incidence rate (IR) and its 95% confidence interval for each treatment group, incidence rate ratio (IRR) of each active MT-7117 treatment group versus placebo, 95% confidence interval of the IRR together

with relevant p-values will be reported.

The following example SAS code will be used;



The percentage of subjects who are responders based on average daily sunlight exposure time to first prodromal symptom associated with sunlight exposure between 1 hour post sunrise and 1 hour pre-sunset defined by within-subject meaningful change of 66 minutes increase from baseline to Week 26, will be analyzed using logistic regression analysis. The model will include the treatment group and the randomization stratification factors as fixed effect and the baseline average daily sunlight exposure time to first prodromal symptom as covariate. The treatment odds ratio at Week 26 will be estimated using a contrast. The missing data at Week 26 due to no available average daily sunlight exposure time to first prodromal symptom will be addressed as non-responder.

For each secondary efficacy endpoint, a subgroup analysis by region (North America, Europe, Japan, Australia) will be done.

#### 8.2.3 Exploratory Efficacy Endpoints

The following exploratory efficacy endpoints will be analysed using the similar model as specified for the primary analysis (MMRM) replacing the baseline average daily sunlight exposure time to first prodromal symptom as covariate with the corresponding covariates at baseline visit in the below bullets.

- Change from baseline in the average daily mean intensity on an 11-point Likert scale of the subject's prodromal symptoms over time during 26-week double-blind treatment period.
- Change from baseline in average daily duration (minutes) of prodromal symptoms during 26-week double-blind treatment period.

- Change from baseline in the average daily mean intensity of the subject's phototoxic reactions (associated with sun exposure) during 26-week double-blind treatment period on an 11-point Likert scale.
- Change from baseline in average daily duration (minutes) of phototoxic reactions (associated with sun exposure) during 26-week double-blind treatment period.
- Change from baseline for all total score and total score in each domain of, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, and pain interference in the PROMIS-57
- Change from baseline in PGIS at each visit.

The following endpoints will be analysed using the same negative binomial model with log link as specified for the secondary efficacy endpoint.

- Total number of sunlight-induced pain events defined as phototoxic events during 26week double-blind treatment.
- Total number of sunlight-induced non-prodrome, phototoxic reactions during 26-week double-blind treatment.

The following endpoint will be analysed using the same logistic regression model as specified for the secondary efficacy endpoint.

• The percentage of subjects who are responders at Week 26 based on PGIC (Very Much Improved or Much Improved).

The following endpoint will be listed and summarized by treatment and planned time point using descriptive statistics. The value of melanin density, change from baseline and % change from baseline in melanin density at each visit by skin segments and average of 6 skin segments will be plotted by treatment. The average of 6 skin segments for the melanin density and for the change from baseline in melanin density at each visit, will be analysed using MMRM model similar to the analyses for the primary endpoint. A subgroup analysis by region (North America, Europe, Japan, Australia), by Fitzpatrick scale test category (I-II or III-VI), by Melanin density at BL (>=Median, <Median) and by the will be done.

• Change from baseline and % change from baseline in melanin density at each visit by skin segments. Average of 6 skin segments for the change from baseline and % change from baseline in melanin density at each visit.

The following endpoints will be analysed using either ANCOVA or ANOVA model. The ANCOVA model will include the treatment group, randomization strata as fixed factors together with continuous covariate terms for the corresponding baseline values except for the below total

time endpoints.

- Change from baseline for in-clinic sunlight exposure time (minutes) to the first prodromal symptoms or end of test, whichever comes first.
- Total time (hours) during the 26-week double-blind treatment period in duration of sunlight exposure between 1 hour post sunrise and 1 hour pre-sunset without prodromal symptoms.
- Total time (hours) during the 26-week double-blind treatment period in duration of sunlight exposure between 1 hour post sunrise and 1 hour pre-sunset without prodromal symptom with the severity of greater than 0 on 11-point Likert scale and without phototoxic reactions (pain-free time hours).
- Change from baseline in average daily duration of sunlight exposure regardless of time of day without prodromal symptoms assessed at Week 26.

The following endpoints will be summarized using descriptive statistics and Wilcoxon's rank sum test.

- Total number of days subject is exposed to sunlight for any duration without prodromal symptoms during 26-week double-blind treatment period.
- Total number of days subject is exposed to sunlight for any duration without prodromal symptom with the severity of greater than 0 on 11-point Likert scale and without phototoxic reactions (pain-free days) during the 26-week double-blind treatment period.
- Total number of days subjects went outdoors during the 26-week double-blind treatment period.
- Total severity of phototoxic reaction on an 11-point Likert scale during the 26-week double-blind treatment period

Maximum severity of photoxic reaction on an 11-point likert scales will be summarized using frequency and percentage. Shift table of maximum phototoxic reaction on an 11-point Likert scale at Week 26 or EOT will be presented using frequency and perenctage.

# For DBE data analysis

All efficacy endpoints in Section 2.3.4 will be simply and descriptively summarized in the ITT2 population in the above similar approach without statistical models.

#### 8.3 Safety Assessments

Safety assessments of DBT period data and DBE period will be made on the SAF1 and SAF2 populations, resepectively. All data will be listed.

#### 8.3.1 Adverse Events

The TEAEs are summarized for subjects with at least one TEAE, at least one treatment emergent adverse event related to study drug, at least one serious TEAE, at least one serious treatment emergent adverse event related to study drug, at least one TEAE leading to drug withdrawal, at least one treatment emergent adverse event related to study drug leading to drug withdrawal, at least one hepatic AE, at least one Adverse Events of Special Interest (AESI) and fatal TEAE. These TEAEs are summarized for subjects by region (North America, Europe, Japan, Australia) as well.

The frequency and incidence of TEAEs will be summarized by System Organ Class (SOC) and Preferred Term (PT) by treatment and overall. For this table, SOC is sorted by International order; then within SOC, PT is sorted by descending counts under MT-7117 group, then descending counts under MT-7117 group, then descending counts under MT-7117 group, then descending counts under Placebo group, then alphabetic order for PTs with the same count.

The AE summaries will be presented for the following:

- TEAEs by SOC and PT
- TEAEs by SOC, PT and severity
- TEAEs by SOC, PT and relationship
- TEAEs by SOC, PT and region (North America, Europe, Japan, Australia)
- Treatment emergent adverse event related to study drugs by SOC and PT
- Treatment emergent adverse event related to study drugs by SOC, PT and severity
- Serious TEAEs by SOC and PT
- Serious treatment emergent adverse event related to study drug s by SOC and PT
- TEAEs leading to drug withdrawn by SOC and PT
- TEAEs by SOC and PT for TEAEs with frequency >= 3% in MT-7117 any treatment groups
- Treatment Emergent Hepatic AEs by SOC and PT
   (Note: Hepatice AE will be defined by SMQ Hepatic List in the appendix)
- AESI by SOC and PT
- TEAEs by SOC, PT and treatment duration
- TEAEs by SOC, PT, treatment duration and region (North America, Europe, Japan, Australia)
- Serious TEAEs by SOC, PT and treatment duration
- TEAEs by SOC and PT (Removing USUBJID: \_\_\_\_\_, \_\_\_\_, \_\_\_\_, \_\_\_\_,

For each of the summaries will be done at the subject level - multiple occurrences of the same event within a subject will be counted once in the summaries by SOC and PT; multiple occurrences of the same event within a subject will be counted once in the maximum intensity category (severe > moderate > mild) and/or maximum drug relationship category (reasonable possibility, no reasonable possibility). If intensity or relationship is found to be missing the most severe occurrence will be imputed for that particular summary.

All AEs for each subject, including multiple occurrences of the same event, will be listed. Deaths that occur during the study will be listed in a data listing. The data listings for serious TEAE and TEAE leading to drug withdrawn will be generated as well.

### 8.3.2 Laboratory Tests

Absolute values and changes from baseline will be summarized for the following laboratory tests parameters. For Haemoglobin, Haematocrit, Red Blood Cell, MCV, Alkaline phosphatase, Aspartate aminotransferase, Alanine aminotransferase, Gamma glutamyl transpeptidase and Bilirubin (direct and total), absolute values and changes from baseline will be summarized by region (North America, Europe, Japan, Australia). Standard Unit will be used for the summary.

| Laboratory Test | Parameters |
|---|---|
| Hematology | Haemoglobin, Haematocrit, Red Blood Cell, Platelet count, MCV, MCH, MCHC, White blood cell count and differential |
| Biochemistry | Alkaline phosphatase, Aspartate aminotransferase, Alanine aminotransferase, Gamma glutamyl transpeptidase, Potassium Sodium, Chloride, Inorganic phosphate, Glucose, Bilirubin (direct and total), Blood urea nitrogen, Cholesterol, Triglycerides, High density lipoprotein cholesterol, Low density lipoprotein cholesterol, Protein (total), Albumin, Creatine kinase, Creatinine, Ferritin, Vitamin D |
| Coagulation | PT, INR, aPTT |
| Urinalysis | Specific gravity, pH, protein, glucose, ketones, urobilinogen, blood Microscopic examination <sup>a</sup> |

<sup>&</sup>lt;sup>a</sup>Performed only if required, based on urinalysis results

Shift table of clinically relevant categories will be presented for the following laboratory tests parameters. The categories will be Low, Normal and High for Hematology, Biochemistry, Urinalysis and Coagulation, and Normal and Abnormal for Urinalysis (Qualitative Value). A shift table of the number and percentage will be provided for subjects who had any post baseline maximum value at any time during the treatment period and met the liver function tests (AST, ALT and Total bilirubin) criteria of the pre-defined limit for the maximum value.

## 8.3.3 Vital Signs

Absolute values and change from baseline will be summarized descriptively and shift table of clinically relevant categories (Normal, Abnormal(Not Clinically Significant, Clinically Significant)) from baseline to EOT will be also presented for the following parameters.

- Systolic Blood Pressure (mmHg)
- Diastolic Blood Pressure (mmHg)
- Pulse Rate
- Respiratory Rate
- Body Temperature (°C)
- Body Weight (kg)

#### 8.3.4 12-Lead ECGs

Absolute values and changes from baseline will be descriptively summarized and shift table of clinically relevant categories (Normal, Abnormal(Not Clinically Significant, Clinically Significant)) from baseline to EOT will be also presented for the following parameters.

- Heart Rate (bpm)
- PR (msec)
- RR (msec)
- QRS (msec)
- QT (msec)
- QTcF (msec)
- QTcB (msec)

A summary table of the number and percentage will be provided for subjects who met the 12-lead ECG criteria of QTcF and QTcB for pre-defined limit as numerator.

#### 8.3.5 Physical Examinations

Physical examination will be summarized with the number and percentage of the subjects for clinically relevant categories (Normal, Abnormal(Not Clinically Significant, Clinically Significant)).

- Abdominal
- Cardiovascular
- General Appearance
- Head
- Eyes
- Ears/nose/throat

- Lymph nodes
- Musculoskeletal
- Neck
- Neurological
- Dermatological
- Other

### 8.3.6 Nevi appearance

Nevi appearance will be summarized with the number and percentage of the subjects' suspicious nevi found:

- Any suspicious nevi found during assessment (Y,N)
- Any clinically significant findings (Y,N).

#### 8.4 Pharmacokinetics Evaluation

Pharmacokinetics evaluation of DBT period data and DBE period will be made on the PK population. All data will be listed.

Plasma concentrations of MT-7117 will be analyzed at randomization visit (pre-dose on Day 1 for not Japanese, 2, 4, 6, and 8 hours post-dose on Day 1 for Japanese), Week 4 (any time), Week 12 (any time), Week 26 (at the visit and 3 to 4 hours after the first PK sample collection), Week 39, (any time) and Week 52 (any time) visits for subjects who are ≥18 to ≤75. For subjects who are ≥12 to ≤17, plasma concentrations of MT-7117 will be analyzed at randomization visit (Day 1, at 2, 4, 6, and 8 hours post-dose), Week 12 (pre-dose and 3 hours post-dose), and Week 26 (pre-dose, 2, and 4 hours post-dose). For the calculation of the summary statistics of palsma concentrations at each sampling point, concentration values reported as below the limit of quantification (BLQ) will be set to 0.

Plasma MT-7117 concentrations will be listed for each subject and scheduled visit and treatment period with the same precision as provided by the bioanalytical laboratory. PK sample collection times, most recent dosing times, as well as derived actual sampling time relative to the most recent dose will be provided in a listing. The actual sampling time relative to the most recent dose will be calculated in hours and rounded to 2 DP.

Plots of individual concentration vs actual sampling time will be presented overlaid with treatment in different symbols for each treatment by visit, or overlaid with visits. Moreover, individual concentrations will be plotted against actual sampling time for each treatment with different symbols for age ( $\geq 12$  to  $\leq 17$  and  $\geq 18$  to  $\leq 75$ ) and ethnicity (Not Japanese and

Japanese) overlaid with visits.

### 8.5 Pharmacogenetics Evaluation

Pharmacogenetics assessments will be made on the ITT1 population.



# 8.6 Exploratory endpoint

Porphyrin and protoporphyrin levels will be listed and summarized using descriptive statistics for the following parameters on the SAF1 and the SAF2 population. Porphyrin and protoporphyrin levels will be summarized by region (North America, Europe, Japan, Australia) as well.

- Plasma total porphyrins(mcg/dL)
- Erythrocyte protoporphyrins(mcg/dL)
- Zinc protoporphyrins(%)
- Metal-Free protoporphyrins(%)

#### 9 DATA PRESENTATION CONVENTIONS

## 9.1 Number of Digits to Report

# (1) Non-PK related

| Statistic . | Specification | Apply to |
|---|---|---|
| Minimum, Maximum | Same number of DPs as<br>the data provided in the<br>datasets | All original (i.e. non-derived) |
| | see section 7.1.2.3 | All derived data |
| Mean, Median, SD, SE,<br>Confidence intervals | One more DP than above | All |
| Percentages*1 | 1 DP | All |

| Ratios | 3 DPs | All |
|------------|-------|-----|
| p-values*2 | 3 DPs | All |

<sup>\*1</sup> Percentages: use 1 place beyond the decimal point, except for the following cases:

If the percentage is equal to 0, then leave blank, do not use (0)

If the percentage is equal to 100, then use "(100)" without a decimal

If the p-value is less than 0.001, then use p<0.001

## (2) PK Plasma Concentration

| Statistic | Specification |
|------------------|----------------------------------------------------------|
| Individual value | 4 significant digits |
| Minimum, Maximum | Same number of DPs as the individual value |
| Mean, SD, Median | Number of DPs securing at least 2 significant digits for |
| | the minimum |

# 9.2 Treatment Groups to Report

| Freatment Group for DRV da | ta analysis For FFLs |
|----------------------------|------------------------|
| MT-7117 | MT-7117 |
| MT-7117 | MT-7117 |
| Placebo | Placebo |

| Incoment Charge | for DBE data analysis | FOR TELS, Marie |
|-----------------|-------------------------|--------------------|
| MT-7117 | | MT-7117 |
| MT-7117 | | MT-7117 |
| MT-7117 | (switched from Placebo) | Placebo -> MT-7117 |
| MT-7117 | (switched from Placebo) | Placebo -> MT-7117 |

## 9.3 Analysis Visits to Report

## eDiary:

| Analysis<br>Visit | Apply to | | | | | |
|---|---|---|---|---|---|---|
| | Analysis | for DBT peri | od data | Analysis for | DBE period da | ta |
| | Change<br>from<br>baseline | Total time / number of days / severity of phototoxic reaction during 26 weeks | Maximum<br>severity of<br>phototoxic<br>reaction | Change<br>from<br>baseline | Total time /<br>number of<br>days /<br>severity of<br>phototoxic<br>reaction<br>during 26<br>weeks | Maximum<br>severity of<br>phototoxic<br>reaction |

<sup>\*2</sup> p-values: use 3 places beyond the decimal point, except for the following cases:

# Statistical Analysis Plan Protocol No. MT-7117-G01

## Mitsubishi Tanabe Pharma Development America

| Baseline | X | <u> </u> | X | | | |
|---|---|---|---|---|---|---|
| Week 2 | X | | 1 | | | |
| Week 4 | X | | | | | |
| Week 6 | X | · | | | | |
| Week 8 | X | , | | ~~~ | | |
| Week 10 | X | | | | | |
| Week 12 | X | | | | | |
| Week 14 | X | | | | | |
| Week 16 | X | | | | | |
| Week 18 | X | | | | | |
| Week 20 | X | | | | | |
| Week 22 | X | | | | | |
| Week 24 | X | | | | | |
| Week 26 | X | | | | | |
| (DBT EOT) | | | | | | |
| During 26 | | X | X | | | X |
| weeks(DBT) | | | | | | |
| EOT for | | | X | | | |
| DBT | | | | | | |
| Follow-up | X | | - | | | |
| until Week | | | | | | |
| 32(DBT | | | | | | |
| EOS) | | | | 37 | | |
| Week 26 | | | | X | 1 | |
| (DBE | | | | | | |
| Baseline) | | | | X | | |
| Week 28 | | | | X | | |
| Week 32 | | | | X | | |
| Week 39<br>Week 52 | | | | X | | X |
| (DBE EOT) | | | | ^ | | ^ |
| During 26 | | | | | X | |
| weeks(DBE) | · | | | | ^ | |
| EOT for | | | | | | |
| DBE | | | | | | |
| Follow-up | | | | X | | |
| until Week | | | | | | |
| 58 (DBE | | | | | | |
| EOS) | | | | | | |

# Efficacy except for eDiary:

| Analysis Apply<br>Visit | / <b>to</b> | in party services | | | |
|---|---|---|---|---|---|
| Analy | sis for DBT | period data | A BOOK TO SERVICE AND A SERVIC | Analysis for | DBE period data |

# Statistical Analysis Plan Protocol No. MT-7117-G01

## Mitsubishi Tanabe Pharma Development America

| | PROMISE | Delo | Heir | | Midami | PROMES. | TRAIC | in Griss | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | 57/ | | | | d pikit | 977 | | | ន្ទាហ៍ស្នែញ | |
| | | | | (1) 10 | evaluation | | | | | a valimitoji k |
| Deseline | v | | v | tësi. | | | | | (i-j) | |
| Baseline | X | 77 | X | X | X | | | | | |
| Week 4 | 37 | X | X | | X | | | | | |
| Week 12 | X | 37 | | 37 | | | | | | |
| Week 26 | X | X | X | X | X | | | | | |
| (DBT | | | | | | | | | | |
| EOT) | 37 | | 37 | | 37 | | | | | |
| Follow- | X | | X | | X | | | | | |
| up until | | | | | | | | | | |
| Week | | | | | | | | | | |
| 32(DBT | | | | | | | | | | |
| EOS) | | | | | | 37 | 37 | 37 | 37 | 77 |
| Week 26 | | | | | | X | X | X | X | X |
| (DBE | | | | | | | | | | İ |
| baseline) | | | | | | v | | X | | |
| Week 39 | | | | | | X | X | X | X | X |
| Week 52 | | | | | | X | A. | X | X | A |
| (DBE | | | | | | | | | | |
| EOT) | | | | | | 37 | | X | | X |
| Follow- | | | | | | X | | A | | ^ |
| up until | | | | | | | | | | |
| Week | | | | | | | | | | |
| 58(DBE | | | | | | | | | | |
| EOS) | | | | | | | | | | |

# Safety:

| Analysis. | Apply to | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Visit 18 | | 1 44 75 52 | 10.786 | | | age to com | de la companya de la companya de la companya de la companya de la companya de la companya de la companya de la | 1.00 |
| | Amalysis for | | | | Analysisio | | | |
| | Eaboratory | E-CHRISTERS BIRT | 30 720 E35 HOUSE REPORT A | THE DEFENDENCE OF STREET | Laboratory | A COLUMN TO A STATE OF THE STATE OF | ENGINEERING CONTRACTOR | A STATE OF THE PARTY OF THE PAR |
| | Tests | Signs | | | Tests 44- | | | evaluation |
| | | | ECGs | | | | ECGs | |
| Screening | X*** | X | | X | | | | |
| Baseline | X*** | X | X | | | | | |
| Week 2 | X (liver function) | | | | | | : | |
| Week 4 | X | X | | X | | | | |
| Week 8 | X (liver function) | | | | | | | |
| Week 12 | X | X | | X | | | | |
| Week 16 | X** | | | | | | | |

| Week 18 | X** | | | Ï | 1 | | · [ · | |
|------------|-----|---|---|---|-----|---|-------|---|
| Week 20 | X** | | | | | | | |
| Week 26 | X | X | X | X | | | | |
| (DBT | | | | | | | | |
| EOT) | | | | | | | | |
| EOT for | X | X | X | X | | | | |
| DBT | | | | | | | | |
| (LOCF) | | | | | | | | |
| Follow-up | X | X | | X | | | | |
| until Week | | | | | | | | |
| 32 (DBT | | | | | | | | |
| EOS) | | | | | | | | |
| Week 26 | | | | | X | X | X | X |
| (DBE | | | | | | | | |
| Baseline) | | | | | | | | |
| Week 28 | | | | | X* | | · | |
| Week 30 | | | | | X** | | | |
| Week 32 | | | | | X* | | | |
| Week 36 | | | | | X** | | | |
| Week 39 | | | | | X | X | | X |
| Week 43 | | | | | X** | | | |
| Week 47 | | | | | X** | | | |
| Week 52 | | | | | X | X | X | X |
| (DBE | | | | | | | | |
| EOT) | | | | | | | | |
| EOT for | | | | | X | X | X | X |
| DBE | | | | | | | | |
| (LOCF) | | | | | | | | |
| Follow-up | | | | | X | X | | X |
| until Week | | | | | | | | |
| 58(DBE | | | | | | | | |
| EOS) | | | | | | | | |

<sup>\*</sup>At Visits 3, 5, 8, and 9, subjects may have mobile units or in-clinic visits to measure liver function markers (ALT, AST, GGT, ALP, direct and total bilirubin). Blood samples for liver function markers will be shipped to the central laboratory.

## 10 CHANGE FROM THE PROTOCOL

There are currently no changes to analysis from protocol.

<sup>\*\*</sup>For only specific country(See Table 4)

<sup>\*\*\*</sup>For liver function markers (ALT, AST, GGT, ALP, direct and total bilirubin), the mean value between a value at screening and at randomization will be treated as a baseline value.

## 11 SOFTWARE

All statistical analyses will be performed using SAS version 9.4 or higher.

## 12 REFERENCES

N/A








# Mitsubishi Tanabe Pharma Development America



## 14 APPENDIX









# Statistical Analysis Plan Protocol No. MT-7117-G01

Mitsubishi Tanabe Pharma Development America



# 14.2 SMQ List of Hepatic TEAE in MedDRA version 23.1

| Bilirubin excretion disorder | 10061009 |
|-----------------------------------------------|----------|
| Cholaemia | 10048611 |
| Cholestasis | 10008635 |
| Cholestatic liver injury | 10067969 |
| Cholestatic pruritus | 10064190 |
| Drug-induced liver injury | 10072268 |
| Hepatitis cholestatic | 10019754 |
| Hyperbilirubinaemia | 10020578 |
| Icterus index increased | 10021209 |
| Jaundice | 10023126 |
| Jaundice cholestatic | 10023129 |
| Jaundice hepatocellular | 10023136 |
| Mixed liver injury | 10066758 |
| Ocular icterus | 10058117 |
| Parenteral nutrition associated liver disease | 10074151 |
| Deficiency of bile secretion | 10071634 |
| Yellow skin | 10048245 |
| Acquired hepatocerebral degeneration | 10080860 |
| Acute hepatic failure | 10000804 |
| Acute on chronic liver failure | 10077305 |
| Acute yellow liver atrophy | 10070815 |
| Ascites | 10003445 |
| Asterixis | 10003547 |
| Bacterascites | 10068547 |
| Biliary cirrhosis | 10004659 |
| Biliary fibrosis | 10004664 |
| Cardiohepatic syndrome | 10082480 |
| Cholestatic liver injury | 10067969 |
| Chronic hepatic failure | 10057573 |
| Coma hepatic | 10010075 |
| Cryptogenic cirrhosis | 10063075 |
| Diabetic hepatopathy | 10071265 |
| Drug-induced liver injury | 10072268 |

| Duodenal varices | 10051010 |
|----------------------------------------------------|----------|
| Flood syndrome | 10084797 |
| Gallbladder varices | 10072319 |
| Gastric variceal injection | 10076237 |
| Gastric variceal ligation | 10076238 |
| Gastric varices | 10051012 |
| Gastric varices haemorrhage | 10057572 |
| Gastrooesophageal variceal haemorrhage prophylaxis | 10066597 |
| Hepatectomy | 10061997 |
| Hepatic atrophy | 10019637 |
| Hepatic calcification | 10065274 |
| Hepatic cirrhosis | 10019641 |
| Hepatic encephalopathy | 10019660 |
| Hepatic encephalopathy prophylaxis | 10066599 |
| Hepatic failure | 10019663 |
| Hepatic fibrosis | 10019668 |
| Hepatic hydrothorax | 10067365 |
| Hepatic infiltration eosinophilic | 10064668 |
| Hepatic lesion | 10061998 |
| Hepatic necrosis | 10019692 |
| Hepatic steato-fibrosis | 10077215 |
| Hepatic steatosis | 10019708 |
| Hepatitis fulminant | 10019772 |
| Hepatobiliary disease | 10062000 |
| Hepatocellular foamy cell syndrome | 10053244 |
| Hepatocellular injury | 10019837 |
| Hepatopulmonary syndrome | 10052274 |
| Hepatorenal failure | 10019845 |
| Hepatorenal syndrome | 10019846 |
| Hepatotoxicity | 10019851 |
| Immune-mediated cholangitis | 10083406 |
| Immune-mediated hepatic disorder | 10083521 |
| Intestinal varices | 10071502 |
| Intestinal varices haemorrhage | 10078058 |
| Liver dialysis | 10076640 |
| Liver disorder | 10024670 |

| Liver injury | 10067125 |
|---------------------------------------|----------|
| Liver operation | 10062040 |
| Liver transplant | 10024714 |
| Lupoid hepatic cirrhosis | 10025129 |
| Minimal hepatic encephalopathy | 10076204 |
| Mixed liver injury | 10066758 |
| Nodular regenerative hyperplasia | 10051081 |
| Nonalcoholic fatty liver disease | 10082249 |
| Non-alcoholic steatohepatitis | 10053219 |
| Non-cirrhotic portal hypertension | 10077259 |
| Oedema due to hepatic disease | 10049631 |
| Oesophageal varices haemorrhage | 10030210 |
| Peripancreatic varices | 10073215 |
| Portal fibrosis | 10074726 |
| Portal hypertension | 10036200 |
| Portal hypertensive colopathy | 10079446 |
| Portal hypertensive enteropathy | 10068923 |
| Portal hypertensive gastropathy | 10050897 |
| Portal vein cavernous transformation | 10073979 |
| Portal vein dilatation | 10073209 |
| Portopulmonary hypertension | 10067281 |
| Primary biliary cholangitis | 10080429 |
| Regenerative siderotic hepatic nodule | 10080679 |
| Renal and liver transplant | 10052279 |
| Retrograde portal vein flow | 10067338 |
| Reye's syndrome | 10039012 |
| Reynold's syndrome | 10070953 |
| Splenic varices | 10067823 |
| Splenic varices haemorrhage | 10068662 |
| Steatohepatitis | 10076331 |
| Subacute hepatic failure | 10056956 |
| Sugiura procedure | 10083010 |
| Varices oesophageal | 10056091 |
| Varicose veins of abdominal wall | 10072284 |
| White nipple sign | 10078438 |
| Anorectal varices | 10068924 |

| Anorectal varices haemorrhage | 10068925 |
|-----------------------------------------------------|----------|
| Complications of transplanted liver | 10010186 |
| Hepatic perfusion disorder | 10083840 |
| Increased liver stiffness | 10082444 |
| Intrahepatic portal hepatic venous fistula | 10072629 |
| Liver and pancreas transplant rejection | 10051603 |
| Liver transplant failure | 10083175 |
| Liver transplant rejection | 10024715 |
| Multivisceral transplantation | 10082450 |
| Peritoneovenous shunt | 10052716 |
| Portal shunt | 10036204 |
| Portal shunt procedure | 10077479 |
| Small-for-size liver syndrome | 10069380 |
| Spider naevus | 10041519 |
| Splenic artery embolisation | 10083795 |
| Splenorenal shunt | 10041661 |
| Splenorenal shunt procedure | 10077281 |
| Spontaneous intrahepatic portosystemic venous shunt | 10076239 |
| Stomal varices | 10075186 |
| Acute graft versus host disease in liver | 10066263 |
| Allergic hepatitis | 10071198 |
| Alloimmune hepatitis | 10080576 |
| Autoimmune hepatitis | 10003827 |
| Chronic graft versus host disease in liver | 10072160 |
| Chronic hepatitis | 10008909 |
| Graft versus host disease in liver | 10064676 |
| Hepatitis | 10019717 |
| Hepatitis acute | 10019727 |
| Hepatitis cholestatic | 10019754 |
| Hepatitis chronic active | 10019755 |
| Hepatitis chronic persistent | 10019759 |
| Hepatitis fulminant | 10019772 |
| Hepatitis toxic | 10019795 |
| Immune-mediated hepatitis | 10078962 |
| Ischaemic hepatitis | 10023025 |
| Lupus hepatitis | 10067737 |

| Non-alcoholic steatohepatitis | 10053219 |
|-----------------------------------------|----------|
| Radiation hepatitis | 10051015 |
| Steatohepatitis | 10076331 |
| Granulomatous liver disease | 10018704 |
| Liver sarcoidosis | 10068664 |
| Portal tract inflammation | 10075331 |
| Benign hepatic neoplasm | 10004269 |
| Benign hepatobiliary neoplasm | 10077922 |
| Focal nodular hyperplasia | 10052285 |
| Haemangioma of liver | 10018821 |
| Haemorrhagic hepatic cyst | 10067796 |
| Hepatic adenoma | 10019629 |
| Hepatic cyst | 10019646 |
| Hepatic cyst ruptured | 10053973 |
| Hepatic haemangioma rupture | 10054885 |
| Hepatic hamartoma | 10079685 |
| Hepatobiliary cyst | 10079889 |
| Cholangiosarcoma | 10077861 |
| Hepatic angiosarcoma | 10067388 |
| Hepatic cancer | 10073069 |
| Hepatic cancer metastatic | 10055110 |
| Hepatic cancer recurrent | 10073070 |
| Hepatic cancer stage I | 10059318 |
| Hepatic cancer stage II | 10059319 |
| Hepatic cancer stage III | 10059324 |
| Hepatic cancer stage IV | 10059325 |
| Hepatobiliary cancer | 10073073 |
| Hepatobiliary cancer in situ | 10073074 |
| Hepatoblastoma | 10062001 |
| Hepatoblastoma recurrent | 10019823 |
| Hepatocellular carcinoma | 10073071 |
| Liver carcinoma ruptured | 10050842 |
| Mixed hepatocellular cholangiocarcinoma | 10027761 |
| Hepatic neoplasm | 10019695 |
| Hepatobiliary neoplasm | 10061203 |
| Alanine aminotransferase abnormal | 10001547 |

| Alanine aminotransferase increased | 10001551 |
|-----------------------------------------------|----------|
| Ammonia abnormal | 10001942 |
| Ammonia increased | 10001946 |
| Ascites | 10003445 |
| Aspartate aminotransferase abnormal | 10003477 |
| Aspartate aminotransferase increased | 10003481 |
| AST/ALT ratio abnormal | 10082832 |
| Bacterascites | 10068547 |
| Bile output abnormal | 10051344 |
| Bile output decreased | 10051343 |
| Biliary ascites | 10074150 |
| Bilirubin conjugated abnormal | 10067718 |
| Bilirubin conjugated increased | 10004685 |
| Bilirubin urine present | 10077356 |
| Biopsy liver abnormal | 10004792 |
| Blood bilirubin abnormal | 10058477 |
| Blood bilirubin increased | 10005364 |
| Blood bilirubin unconjugated increased | 10005370 |
| Bromosulphthalein test abnormal | 10006408 |
| Child-Pugh-Turcotte score abnormal | 10077020 |
| Child-Pugh-Turcotte score increased | 10068287 |
| Computerised tomogram liver abnormal | 10078360 |
| Congestive hepatopathy | 10084058 |
| Foetor hepaticus | 10052554 |
| Galactose elimination capacity test abnormal | 10059710 |
| Galactose elimination capacity test decreased | 10059712 |
| Gamma-glutamyltransferase abnormal | 10017688 |
| Gamma-glutamyltransferase increased | 10017693 |
| Guanase increased | 10051333 |
| Hepaplastin abnormal | 10019621 |
| Hepaplastin decreased | 10019622 |
| Hepatic artery flow decreased | 10068997 |
| Hepatic enzyme abnormal | 10062685 |
| Hepatic enzyme decreased | 10060794 |
| Hepatic enzyme increased | 10060795 |
| Hepatic function abnormal | 10019670 |

| Hepatic hyperfusion 10076254 Hepatic hypoperfusion 10084751 Hepatic mass 10057110 Hepatic pain 10019705 Hepatic sequestration 10066244 Hepatic vascular resistance increased 10068358 Hepatic venous pressure gradient abnormal 10083172 Hepatic venous pressure gradient increased 10083171 Hepatobiliary scan abnormal 10066195 Hepatomegaly 10019842 Hepatosplenomegaly 10019847 Hyperammonaemia 10020575 Hyperbilirubinaemia 10020575 Hyperbolia 10051924 Hypertransaminasaemia 10068237 Kayser-Fleischer ring 10023321 Liver function test abnormal 10024502 Liver function test decreased 10077677 Liver function test increased 10077672 Liver palpable 10075895 Liver rederness 10061947 Liver rederness 10061947 Magnetic resonance imaging liver abnormal 10082443 Mitochondrial aspartate aminotransferase increased | Hepatic hydrothorax | 10067365 |
|---|---|---|
| Hepatic mass 10057110 Hepatic pain 10019705 Hepatic sequestration 10066244 Hepatic vascular resistance increased 1006358 Hepatic venous pressure gradient abnormal 10083172 Hepatic venous pressure gradient increased 10083171 Hepatobiliary scan abnormal 10066195 Hepatomegaly 10019842 Hepatosplenomegaly 10019847 Hyperammonaemia 10020575 Hyperbilirubinaemia 10020578 Hyperbilirubinaemia 10020578 Hypertransaminasaemia 10068237 Kayser-Fleischer ring 10023321 Liver function test abnormal 10024690 Liver function test decreased 10077677 Liver function test increased 10077672 Liver function test increased 100752550 Liver palpable 10075895 Liver tenderness 10024712 Magnetic resonance imaging liver abnormal 10061947 Liver tenderness 10024712 Magnetic resonance proton density fat fraction measurement 1008243 <t< td=""><td>Hepatic hypertrophy</td><td>10076254</td></t<> | Hepatic hypertrophy | 10076254 |
| Hepatic pain 10019705 Hepatic sequestration 10066244 Hepatic vascular resistance increased 10068358 Hepatic venous pressure gradient abnormal 10083172 Hepatic venous pressure gradient increased 10083171 Hepatobiliary scan abnormal 10066195 Hepatomegaly 10019842 Hepatomegaly 10019847 Hyperammonaemia 10020575 Hyperbilirubinaemia 10020578 Hyperbilirubinaemia 10020578 Hypertansaminasaemia 10068237 Kayser-Fleischer ring 10023321 Liver function test abnormal 10024690 Liver function test decreased 10077677 Liver function test increased 10077692 Liver induration 10052550 Liver palpable 10075895 Liver scan abnormal 10061947 Liver tendemess 10024712 Magnetic resonance imaging liver abnormal 10083123 Magnetic resonance proton density fat fraction measurement 10082443 Mitochondrial aspartate aminotransferase increased 10074712 Molar ratio of total branched-chain amino acid to tyrosine 10066869 Oedema due to hepatic disease 10049631 Perihepatic discomfort 10054125 Retrograde portal vein flow 10067338 Transaminases increased 10045428 Ultrasound liver abnormal 10062688 Ultrasound liver abnormal 10045428 Ultrasound liver abn | Hepatic hypoperfusion | 10084751 |
| Hepatic sequestration | Hepatic mass | 10057110 |
| Hepatic vascular resistance increased 10068358 Hepatic venous pressure gradient abnormal 10083172 Hepatic venous pressure gradient increased 10083171 Hepatobiliary scan abnormal 10066195 Hepatomegaly 10019842 Hepatosplenomegaly 10019847 Hyperammonaemia 10020575 Hyperbilirubinaemia 10020578 Hypercholia 10051924 Hypertransaminasaemia 10068237 Kayser-Fleischer ring 10023321 Liver function test abnormal 10024690 Liver function test decreased 10077677 Liver function test increased 10077692 Liver induration 10052550 Liver palpable 10075895 Liver scan abnormal 10061947 Liver tenderness 10024712 Magnetic resonance imaging liver abnormal 10083123 Magnetic resonance proton density fat fraction measurement 10082443 Mitochondrial aspartate aminotransferase increased 10064712 Molar ratio of total branched-chain amino acid to tyrosine 10066869 Oedema due to h | Hepatic pain | 10019705 |
| Hepatic venous pressure gradient abnormal 10083172 Hepatic venous pressure gradient increased 10083171 Hepatobiliary scan abnormal 1006195 Hepatomegaly 10019842 Hepatosplenomegaly 10019847 Hyperammonaemia 10020575 Hyperbilirubinaemia 10020578 Hypercholia 10051924 Hypertransaminasaemia 10068237 Kayser-Fleischer ring 10023321 Liver function test abnormal 10024690 Liver function test decreased 10077677 Liver function test increased 10077692 Liver induration 10052550 Liver palpable 10075895 Liver scan abnormal 10061947 Liver tenderness 10024712 Magnetic resonance imaging liver abnormal 10083123 Magnetic resonance proton density fat fraction measurement 1008243 Mitochondrial aspartate aminotransferase increased 10064712 Molar ratio of total branched-chain amino acid to tyrosine 10066869 Oedema due to hepatic disease 10049631 Perihepatic discomfort <td>Hepatic sequestration</td> <td>10066244</td> | Hepatic sequestration | 10066244 |
| Hepatic venous pressure gradient increased 10083171 Hepatobiliary scan abnormal 10066195 Hepatomegaly 10019842 Hepatosplenomegaly 10019847 Hyperammonaemia 10020575 Hyperbilirubinaemia 10020578 Hypercholia 10051924 Hypertransaminasaemia 10068237 Kayser-Fleischer ring 10023321 Liver function test abnormal 10024690 Liver function test decreased 10077677 Liver function test increased 10077692 Liver induration 10052550 Liver palpable 10075895 Liver scan abnormal 10061947 Liver tenderness 10024712 Magnetic resonance imaging liver abnormal 10083123 Magnetic resonance proton density fat fraction measurement 10082443 Mitochondrial aspartate aminotransferase increased 10064712 Molar ratio of total branched-chain amino acid to tyrosine 10066869 Oedema due to hepatic disease 10049631 Perihepatic discomfort 10054125 Retrograde portal vein flow < | Hepatic vascular resistance increased | 10068358 |
| Hepatobiliary scan abnormal 10066195 Hepatomegaly 10019842 Hepatosplenomegaly 10019847 Hyperammonaemia 10020575 Hyperbilirubinaemia 10020578 Hypercholia 10051924 Hypertransaminasaemia 10068237 Kayser-Fleischer ring 10023321 Liver function test abnormal 10024690 Liver function test decreased 10077677 Liver function test increased 10077692 Liver induration 10052550 Liver palpable 10075895 Liver scan abnormal 10061947 Liver tenderness 10024712 Magnetic resonance imaging liver abnormal 10083123 Magnetic resonance proton density fat fraction measurement 10082443 Mitochondrial aspartate aminotransferase increased 10064712 Molar ratio of total branched-chain amino acid to tyrosine 10066869 Oedema due to hepatic disease 10049631 Perihepatic discomfort 10054125 Retrograde portal vein flow 10067338 Total bile acids increased 10064558 | Hepatic venous pressure gradient abnormal | 10083172 |
| Hepatosplenomegaly 10019847 Hyperammonaemia 10020575 Hyperbilirubinaemia 10020578 Hypercholia 10051924 Hypertransaminasaemia 10068237 Kayser-Fleischer ring 10023321 Liver function test abnormal 10024690 Liver function test decreased 10077677 Liver function test increased 10077692 Liver induration 10052550 Liver palpable 10075895 Liver scan abnormal 10061947 Liver tenderness 10024712 Magnetic resonance imaging liver abnormal 10083123 Magnetic resonance proton density fat fraction measurement 10082443 Mitochondrial aspartate aminotransferase increased 10064712 Molar ratio of total branched-chain amino acid to tyrosine 10066869 Oedema due to hepatic disease 10049631 Perihepatic discomfort 10054125 Retrograde portal vein flow 10067338 Total bile acids increased 10064558 Transaminases abnormal 10062688 Transaminases increased 1005488 | Hepatic venous pressure gradient increased | 10083171 |
| Hepatosplenomegaly 10019847 Hyperammonaemia 10020575 Hyperbilirubinaemia 10020578 Hypercholia 10051924 Hypertransaminasaemia 10068237 Kayser-Fleischer ring 10023321 Liver function test abnormal 10024690 Liver function test decreased 10077677 Liver function test increased 10077692 Liver induration 10052550 Liver palpable 10075895 Liver scan abnormal 10061947 Liver tenderness 10024712 Magnetic resonance imaging liver abnormal 10083123 Magnetic resonance proton density fat fraction measurement 10082443 Mitochondrial aspartate aminotransferase increased 10064712 Molar ratio of total branched-chain amino acid to tyrosine 10066869 Oedema due to hepatic disease 10049631 Perihepatic discomfort 10054125 Retrograde portal vein flow 10067338 Total bile acids increased 10064558 Transaminases abnormal 10062688 Transaminases increased 1005488 | Hepatobiliary scan abnormal | 10066195 |
| Hyperammonaemia 10020575 Hyperbilirubinaemia 10020578 Hypercholia 10051924 Hypertransaminasaemia 10068237 Kayser-Fleischer ring 10023321 Liver function test abnormal 10024690 Liver function test decreased 10077677 Liver function test increased 10077692 Liver induration 10052550 Liver palpable 10075895 Liver scan abnormal 10061947 Liver tenderness 10024712 Magnetic resonance imaging liver abnormal 10083123 Magnetic resonance proton density fat fraction measurement 10082443 Mitochondrial aspartate aminotransferase increased 10064712 Molar ratio of total branched-chain amino acid to tyrosine 10066869 Oedema due to hepatic disease 10049631 Perihepatic discomfort 10054125 Retrograde portal vein flow 10067338 Total bile acids increased 10064558 Transaminases abnormal 10062688 Transaminases increased 10054889 Ultrasound liver abnormal 10045428 | Hepatomegaly | 10019842 |
| Hyperbilirubinaemia 10020578 Hypercholia 10051924 Hypertransaminasaemia 10068237 Kayser-Fleischer ring 10023321 Liver function test abnormal 10024690 Liver function test decreased 10077677 Liver function test increased 10077692 Liver induration 10052550 Liver palpable 10075895 Liver scan abnormal 10061947 Liver tenderness 10024712 Magnetic resonance imaging liver abnormal 10083123 Magnetic resonance proton density fat fraction measurement 10082443 Mitochondrial aspartate aminotransferase increased 10064712 Molar ratio of total branched-chain amino acid to tyrosine 10066869 Oedema due to hepatic disease 10049631 Perihepatic discomfort 10054125 Retrograde portal vein flow 10067338 Total bile acids increased 10064558 Transaminases abnormal 10062688 Transaminases increased 10054889 Ultrasound liver abnormal 10045428 | Hepatosplenomegaly | 10019847 |
| Hypercholia 10051924 Hypertransaminasaemia 10068237 Kayser-Fleischer ring 10023321 Liver function test abnormal 10024690 Liver function test decreased 10077677 Liver function test increased 10077692 Liver induration 10052550 Liver palpable 10075895 Liver scan abnormal 10061947 Liver tenderness 10024712 Magnetic resonance imaging liver abnormal 10083123 Magnetic resonance proton density fat fraction measurement 10082443 Mitochondrial aspartate aminotransferase increased 10064712 Molar ratio of total branched-chain amino acid to tyrosine 10066869 Oedema due to hepatic disease 10049631 Perihepatic discomfort 10054125 Retrograde portal vein flow 10067338 Total bile acids increased 10064558 Transaminases abnormal 10062688 Transaminases increased 10054889 Ultrasound liver abnormal 10045428 | Hyperammonaemia | 10020575 |
| Hypertransaminasaemia 10068237 Kayser-Fleischer ring 10023321 Liver function test abnormal 10024690 Liver function test decreased 10077677 Liver function test increased 10077692 Liver induration 10052550 Liver palpable 10075895 Liver scan abnormal 10061947 Liver tenderness 10024712 Magnetic resonance imaging liver abnormal 10083123 Magnetic resonance proton density fat fraction measurement 10082443 Mitochondrial aspartate aminotransferase increased 10064712 Molar ratio of total branched-chain amino acid to tyrosine 10066869 Oedema due to hepatic disease 10049631 Perihepatic discomfort 10054125 Retrograde portal vein flow 10067338 Total bile acids increased 10064588 Transaminases abnormal 10062688 Transaminases increased 10054889 Ultrasound liver abnormal 10045428 | Hyperbilirubinaemia | 10020578 |
| Kayser-Fleischer ring10023321Liver function test abnormal10024690Liver function test decreased10077677Liver function test increased10077692Liver induration10052550Liver palpable10075895Liver scan abnormal10061947Liver tenderness10024712Magnetic resonance imaging liver abnormal10083123Magnetic resonance proton density fat fraction measurement10082443Mitochondrial aspartate aminotransferase increased10064712Molar ratio of total branched-chain amino acid to tyrosine10066869Oedema due to hepatic disease10049631Perihepatic discomfort10054125Retrograde portal vein flow10067338Total bile acids increased10064558Transaminases abnormal10062688Transaminases increased10054889Ultrasound liver abnormal10045428 | Hypercholia | 10051924 |
| Liver function test abnormal Liver function test decreased 10077677 Liver function test increased 10077692 Liver induration 10052550 Liver palpable 10075895 Liver scan abnormal 10061947 Liver tenderness 10024712 Magnetic resonance imaging liver abnormal 10083123 Magnetic resonance proton density fat fraction measurement 10082443 Mitochondrial aspartate aminotransferase increased 10064712 Molar ratio of total branched-chain amino acid to tyrosine 10066869 Oedema due to hepatic disease 10049631 Perihepatic discomfort 10054125 Retrograde portal vein flow 10067338 Total bile acids increased 10064558 Transaminases abnormal 10062688 Transaminases increased 10054889 Ultrasound liver abnormal 10045428 | Hypertransaminasaemia | 10068237 |
| Liver function test decreased 10077677 Liver function test increased 10077692 Liver induration 10052550 Liver palpable 10075895 Liver scan abnormal 10061947 Liver tenderness 10024712 Magnetic resonance imaging liver abnormal 10083123 Magnetic resonance proton density fat fraction measurement 10082443 Mitochondrial aspartate aminotransferase increased 10064712 Molar ratio of total branched-chain amino acid to tyrosine 10066869 Oedema due to hepatic disease 10049631 Perihepatic discomfort 10054125 Retrograde portal vein flow 10067338 Total bile acids increased 10064558 Transaminases abnormal 10062688 Transaminases increased 10054889 Ultrasound liver abnormal 10045428 | Kayser-Fleischer ring | 10023321 |
| Liver function test increased 10077692 Liver induration 10052550 Liver palpable 10075895 Liver scan abnormal 10061947 Liver tenderness 10024712 Magnetic resonance imaging liver abnormal 10083123 Magnetic resonance proton density fat fraction measurement 10082443 Mitochondrial aspartate aminotransferase increased 10064712 Molar ratio of total branched-chain amino acid to tyrosine 10066869 Oedema due to hepatic disease 10049631 Perihepatic discomfort 10054125 Retrograde portal vein flow 10067338 Total bile acids increased 10064558 Transaminases abnormal 10062688 Transaminases increased 10054889 Ultrasound liver abnormal 10045428 | Liver function test abnormal | 10024690 |
| Liver induration 10052550 Liver palpable 10075895 Liver scan abnormal 10061947 Liver tenderness 10024712 Magnetic resonance imaging liver abnormal 10083123 Magnetic resonance proton density fat fraction measurement 10082443 Mitochondrial aspartate aminotransferase increased 10064712 Molar ratio of total branched-chain amino acid to tyrosine 10066869 Oedema due to hepatic disease 10049631 Perihepatic discomfort 10054125 Retrograde portal vein flow 10067338 Total bile acids increased 10064558 Transaminases abnormal 10062688 Transaminases increased 10054889 Ultrasound liver abnormal 10045428 | Liver function test decreased | 10077677 |
| Liver palpable 10075895 Liver scan abnormal 10061947 Liver tenderness 10024712 Magnetic resonance imaging liver abnormal 10083123 Magnetic resonance proton density fat fraction measurement 10082443 Mitochondrial aspartate aminotransferase increased 10064712 Molar ratio of total branched-chain amino acid to tyrosine 10066869 Oedema due to hepatic disease 10049631 Perihepatic discomfort 10054125 Retrograde portal vein flow 10067338 Total bile acids increased 10064558 Transaminases abnormal 10062688 Transaminases increased 10054889 Ultrasound liver abnormal 10045428 | Liver function test increased | 10077692 |
| Liver scan abnormal 10061947 Liver tenderness 10024712 Magnetic resonance imaging liver abnormal 10083123 Magnetic resonance proton density fat fraction measurement 10082443 Mitochondrial aspartate aminotransferase increased 10064712 Molar ratio of total branched-chain amino acid to tyrosine 10066869 Oedema due to hepatic disease 10049631 Perihepatic discomfort 10054125 Retrograde portal vein flow 10067338 Total bile acids increased 10064558 Transaminases abnormal 10062688 Transaminases increased 10054889 Ultrasound liver abnormal 10045428 | Liver induration | 10052550 |
| Liver tenderness 10024712 Magnetic resonance imaging liver abnormal 10083123 Magnetic resonance proton density fat fraction measurement 10082443 Mitochondrial aspartate aminotransferase increased 10064712 Molar ratio of total branched-chain amino acid to tyrosine 10066869 Oedema due to hepatic disease 10049631 Perihepatic discomfort 10054125 Retrograde portal vein flow 10067338 Total bile acids increased 10064558 Transaminases abnormal 10062688 Transaminases increased 10054889 Ultrasound liver abnormal 10045428 | Liver palpable | 10075895 |
| Magnetic resonance imaging liver abnormal10083123Magnetic resonance proton density fat fraction measurement10082443Mitochondrial aspartate aminotransferase increased10064712Molar ratio of total branched-chain amino acid to tyrosine10066869Oedema due to hepatic disease10049631Perihepatic discomfort10054125Retrograde portal vein flow10067338Total bile acids increased10064558Transaminases abnormal10062688Transaminases increased10054889Ultrasound liver abnormal10045428 | Liver scan abnormal | 10061947 |
| Magnetic resonance proton density fat fraction measurement Mitochondrial aspartate aminotransferase increased Molar ratio of total branched-chain amino acid to tyrosine Oedema due to hepatic disease Perihepatic discomfort Retrograde portal vein flow Total bile acids increased Transaminases abnormal Ultrasound liver abnormal 10082443 10064712 10066869 10066869 100649631 10067338 10067338 10067338 10062688 | Liver tenderness | 10024712 |
| Mitochondrial aspartate aminotransferase increased 10064712 Molar ratio of total branched-chain amino acid to tyrosine 10066869 Oedema due to hepatic disease 10049631 Perihepatic discomfort 10054125 Retrograde portal vein flow 10067338 Total bile acids increased 10064558 Transaminases abnormal 10062688 Transaminases increased 10054889 Ultrasound liver abnormal 10045428 | Magnetic resonance imaging liver abnormal | 10083123 |
| Molar ratio of total branched-chain amino acid to tyrosine10066869Oedema due to hepatic disease10049631Perihepatic discomfort10054125Retrograde portal vein flow10067338Total bile acids increased10064558Transaminases abnormal10062688Transaminases increased10054889Ultrasound liver abnormal10045428 | Magnetic resonance proton density fat fraction measurement | 10082443 |
| Oedema due to hepatic disease10049631Perihepatic discomfort10054125Retrograde portal vein flow10067338Total bile acids increased10064558Transaminases abnormal10062688Transaminases increased10054889Ultrasound liver abnormal10045428 | Mitochondrial aspartate aminotransferase increased | 10064712 |
| Perihepatic discomfort10054125Retrograde portal vein flow10067338Total bile acids increased10064558Transaminases abnormal10062688Transaminases increased10054889Ultrasound liver abnormal10045428 | Molar ratio of total branched-chain amino acid to tyrosine | 10066869 |
| Retrograde portal vein flow10067338Total bile acids increased10064558Transaminases abnormal10062688Transaminases increased10054889Ultrasound liver abnormal10045428 | Oedema due to hepatic disease | 10049631 |
| Total bile acids increased 10064558 Transaminases abnormal 10062688 Transaminases increased 10054889 Ultrasound liver abnormal 10045428 | Perihepatic discomfort | 10054125 |
| Transaminases abnormal10062688Transaminases increased10054889Ultrasound liver abnormal10045428 | Retrograde portal vein flow | 10067338 |
| Transaminases increased 10054889 Ultrasound liver abnormal 10045428 | Total bile acids increased | 10064558 |
| Ultrasound liver abnormal 10045428 | Transaminases abnormal | 10062688 |
| | Transaminases increased | 10054889 |
| Urine bilirubin increased 10050792 | Ultrasound liver abnormal | 10045428 |
| | Urine bilirubin increased | 10050792 |

| White nipple sign | 10078438 |
|---------------------------------------------------|----------|
| X-ray hepatobiliary abnormal | 10056536 |
| 5'nucleotidase increased | 10000028 |
| AST to platelet ratio index increased | 10084175 |
| Blood alkaline phosphatase abnormal | 10059571 |
| Blood alkaline phosphatase increased | 10059570 |
| Blood cholinesterase abnormal | 10005429 |
| Blood cholinesterase decreased | 10005430 |
| Deficiency of bile secretion | 10071634 |
| Glutamate dehydrogenase increased | 10049483 |
| Glycocholic acid increased | 10080824 |
| Haemorrhagic ascites | 10059766 |
| Hepatic fibrosis marker abnormal | 10074084 |
| Hepatic fibrosis marker increased | 10074413 |
| Hepatic lymphocytic infiltration | 10079686 |
| Hypoalbuninaemia | 10020942 |
| Leucine aminopeptidase increased | 10024275 |
| Liver iron concentration abnormal | 10074352 |
| Liver iron concentration increased | 10074354 |
| Liver opacity | 10084071 |
| Model for end stage liver disease score abnormal | 10077291 |
| Model for end stage liver disease score increased | 10077292 |
| Periportal oedema | 10068821 |
| Peritoneal fluid protein abnormal | 10069000 |
| Peritoneal fluid protein decreased | 10068999 |
| Peritoneal fluid protein increased | 10068998 |
| Pneumobilia | 10066004 |
| Portal vein flow decreased | 10067337 |
| Portal vein pressure increased | 10064936 |
| Retinol binding protein decreased | 10048473 |
| Urobilinogen urine decreased | 10070480 |
| Urobilinogen urine increased | 10070479 |
| Acquired antithrombin III deficiency | 10074561 |
| Acquired factor IX deficiency | 10082747 |
| Acquired factor VIII deficiency | 10082745 |
| Acquired factor XI deficiency | 10082746 |

| Acquired protein S deficiency | 10068370 |
|------------------------------------------|----------|
| Anti factor X activity abnormal | 10077670 |
| Anti factor X activity decreased | 10077674 |
| Anti factor X activity increased | 10077671 |
| Antithrombin III decreased | 10049547 |
| Blood fibrinogen abnormal | 10005518 |
| Blood fibrinogen decreased | 10005520 |
| Blood thrombin abnormal | 10005818 |
| Blood thrombin decreased | 10005820 |
| Blood thromboplastin abnormal | 10005824 |
| Blood thromboplastin decreased | 10005826 |
| Coagulation factor decreased | 10009736 |
| Coagulation factor IX level abnormal | 10061770 |
| Coagulation factor IX level decreased | 10009746 |
| Coagulation factor V level abnormal | 10061771 |
| Coagulation factor V level decreased | 10009754 |
| Coagulation factor VII level abnormal | 10061772 |
| Coagulation factor VII level decreased | 10009761 |
| Coagulation factor X level abnormal | 10061774 |
| Coagulation factor X level decreased | 10009775 |
| Hyperfibrinolysis | 10074737 |
| Hypocoagulable state | 10020973 |
| Hypofibrinogenaemia | 10051125 |
| Hypoprothrombinaemia | 10021085 |
| Hypothrombinaemia | 10058517 |
| Hypothromboplastinaemia | 10058518 |
| International normalised ratio abnormal | 10022592 |
| International normalised ratio increased | 10022595 |
| Protein C decreased | 10037005 |
| Protein S abnormal | 10051736 |
| Protein S decreased | 10051120 |
| Prothrombin level abnormal | 10037048 |
| Prothrombin level decreased | 10037050 |
| Prothrombin time abnormal | 10037057 |
| Prothrombin time prolonged | 10037063 |
| Prothrombin time ratio abnormal | 10061918 |

Statistical Analysis Plan Protocol No. MT-7117-G01

# Mitsubishi Tanabe Pharma Development America

| Prothrombin time ratio increased | <br>10037068 |
|----------------------------------|--------------|
| Thrombin time abnormal | <br>10051319 |
| Thrombin time prolonged | 10051390 |